# Zonisamide/Bupropion Effects on Switching to Electronic Cigarettes (BuZonE)

NCT04388319

Protocol V3.0 16 Feb 2021



Main Office • 7920 ACC Blvd., Suite 110 • Raleigh, NC 27617

**Clinical Study Protocol** 

**Study Title:** Zonisamide/bupropion effects on Switching to Electronic

Cigarettes

**Sponsor:** Foundation for a Smoke-Free World

**Version Number:** Version 3.0

**Version Date:** February 16, 2021

**Principal Investigator:** Jed E. Rose, Ph.D.

Medical Supervision: Perry Willette, MD

**Authors:** Jed E. Rose, Ph.D.,

President and CEO,

Rose Research Center

Perry Willette, MD Medical Director,

Rose Research Center

Tanaia Loeback

Executive Vice President, Rose Research Center

**David Botts** 

Executive Vice President, Rose Research Center

Data and information contained in this document are considered to constitute trade secrets and confidential commercial information, and the legal protections provided to such trade secrets and confidential information are hereby claimed under the applicable provisions of United States law. No part of this document may be publicly disclosed without the written consent of the Rose Research Center, LLC.

# TABLE OF CONTENTS

| Lis | st of Ab | breviationsbreviations | 5 |
|-----|----------|------------------------------------------------------|------|
| 1 | Intro | oduction | 7 |
| | 1.1 | Study Design and Plan | 7 |
| | 1.2 | Background | 7 |
| 2 | Stud | ly Objectives and Endpoints | 8 |
| | 2.1 | Complete Switching from CC to Halo G6 | 8 |
| | 2.2 | Point Abstinence (From CC) at Six Months Post Switch | 8 |
| | 2.3 | Change in Rewarding Effects of Smoking Cigarettes | 8 |
| 3 | Inve | stigational Plan | 8 |
| | 3.1 | Overall Study Design and Plan | 8 |
| | 3.2 | Study Procedures | 9 |
| | 3.3 | Point of Enrollment | . 10 |
| | 3.4 | Study and Session Durations | . 10 |
| 4 | Part | icipant Involvement | 10 |
| | 4.1 | Selection of Study Population | . 10 |
| | 4.2 | Recruitment Strategies | . 12 |
| | 4.3 | Participant Retention in the Study | . 12 |
| | 4.4 | Discontinuation of Participants from Study | . 12 |
| | 4.5 | Lost to Follow-up | . 13 |
| | 4.6 | Violation of Inclusion/Exclusion Criteria | . 13 |
| | 4.7 | Participant Compensation | . 13 |
| | 4.8 | Session and Response Windows | . 13 |
| 5 | Halo | o-G6 Electronic Nicotine Delivery System | 14 |
| | 5.1 | Description of Halo G6 | . 14 |
| | 5.2 | Description of E-Liquid | . 14 |
| | 5.3 | Product Use Timeframe | . 14 |
| | 5.4 | Accountability and Compliance | . 14 |
| 6 | Zoni | samide | 15 |
| | 6.1 | Description of Zonisamide | . 15 |
| | 6.2 | Dosage | . 15 |
| | 6.3 | Dose Adjustment Procedures | . 15 |

| | 6.4 | Accountability and Compliance | 15 |
|----|-------|-----------------------------------------------------|----|
| 7 | Bup | ropion | 16 |
| | 7.1 | Description of Bupropion | 16 |
| | 7.2 | Dosage | 16 |
| | 7.3 | Dose Adjustment Procedures | 16 |
| | 7.4 | Accountability and Compliance | 16 |
| 8 | Stuc | ly Procedures and Activities | 17 |
| | 8.1 | Informed Consent and Guidance | 17 |
| | 8.2 | Safety Laboratory and Other Assessments | 17 |
| | 8.3 | 5-Day Smoking Baseline Collection | 22 |
| | 8.4 | 6-Month Follow Up | 22 |
| | 8.5 | Schedule of Events | 23 |
| | 8.6 | SMS Messaging | 24 |
| 9 | Risk | / Benefit Information | 24 |
| | 9.1 | Potential Risks | 24 |
| | 9.2 | Protection Against Risks | 25 |
| 10 | ) Qua | lity Control and Quality Assurance | 26 |
| | 10.1 | Training of Staff | 26 |
| | 10.2 | Audits and Inspections | 26 |
| 11 | . Rep | orting of Adverse Events | 26 |
| | 11.1 | Definitions | 26 |
| | 11.2 | Collection of Safety Events from Participants | 27 |
| | 11.3 | Assessment of Adverse Events | 28 |
| | 11.4 | Follow-up of Non-serious and Serious Adverse Events | 28 |
| | 11.5 | Reporting of Safety Events to IRB | 29 |
| | 11.6 | Reporting of Safety Events to FDA | 29 |
| | 11.7 | Reporting and Follow-Up of Pregnancies | 29 |
| | 11.8 | Adverse Event Leading to Discontinuation | 29 |
| 12 | Data | Management | 29 |
| | 12.1 | Data Collection Procedures | 29 |
| | 12.2 | Protocol Deviations / Noncompliance | 30 |
| | 12.3 | Data Capture | |
| | 12.4 | Data Handling | 31 |

| 13 Pla | nned Statistical Methods | 31 |
|---|---|---|
| 13.1 | Outcomes | 31 |
| 13.2 | Interim Analysis | 31 |
| 14 Eth | nics and Regulations | 31 |
| 14.1 | IRB Approval | 31 |
| 14.2 | Investigational New Drug Application | |
| 14.3 | Investigational Tobacco Product Application | |
| | • | |
| 14.4 | GCP and Regulatory Requirements | |
| 14.5 | Participant Information and Consent | 32 |
| 14.6 | Amendment to Informed Consent Form | 32 |
| 15 Ad | ministrative Considerations | 33 |
| 15.1 | Participant Confidentiality | 33 |
| 15.2 | Record Retention | 33 |
| | ferences | |
| APPEI | | |
| | ix 1 - Patient Health Questionnaire (PHQ-9) | |
| | ix 2 – Fagerström Test for Nicotine Dependence (FTND) | |
| | ix 3 - Research Participant Payment Verification Form | |
| • • | ix 4 – Smoking History | |
| | ix 5 – Registration Form | |
| • • | ix 6 – Medical History Formix 7- Review of Systems Form | |
| | ix 8 – Employment History | |
| | ix 9 – modified Cigarette Evaluation Questionnaire - Ext (mCEQ-E) | |
| | ix 10 – modified Electronic Cigarette Evaluation Questionnaire - Ext (mECEQ-E) | |
| | ix 11 – Halo G6 Flavor Assessment Questionnaire | |
| Append | ix 12 – Participant Instructions for Varenicline | 55 |
| Append | ix 13 – Participant Instructions for Zonisamide | 56 |
| | ix 14 – Assessment of Behavioral OUTcomes (ABOUT) | |
| Append | ix 15 – Session Payment Form | 59 |
| • • | ix 16 – Reasons to Smoke | |
| Append | ix 17 — Shiffman Jarvik Withdrawal Scale | 61 |

# LIST OF ABBREVIATIONS

AE Adverse event

ALT Alanine aminotransferase

AP Alkaline phosphatase

ASP Application Service Provider

AST Aspartate aminotransferase

BUN Blood urea nitrogen

CC Conventional cigarette

CDC Center for Disease Control and Prevention

CFR Code of Federal Regulations

CO Carbon monoxide

CRF Case report form

CRM Customer relationship management

ECG Electrocardiogram

EOS End of Study

FDA Food and Drug Administration

FTND Fagerström test for nicotine dependence

GCP Good Clinical Practice

HCG Human chorionic gonadotropin

ICF Informed consent form

ICH International Conference on Harmonisation

IRB Institutional Review Board

Kg Kilograms

Lbs pounds

QTc Corrected QT interval

mCEQ Modified Cigarette Evaluation Questionnaire.

MCH Mean corpuscular hemoglobin

MCHC Mean corpuscular hemoglobin concentration

MCV Mean corpuscular volume

Mg Milligram

mL Milliliter

MNWS Minnesota Nicotine Withdrawal Scale

PHQ-9 The Patient Health Questionnaire

PPM Parts per million

RBC Red blood cell

RCT Randomized Control Trial

RRC Rose Research Center, LLC.

SaaS Software-as-a-Service

SAE Serious adverse event

SMS Short Message Service

SOP Standard operating procedure

SSL Secure Sockets Layer

STAI State-Trait Anxiety Inventory

TLS Transport Layer Security

WBC White blood cell

WHO World Health Organization

WI-PREPARE The Wisconsin Predicting Patients' Relapse Questionnaire

# 1 Introduction

#### 1.1 STUDY DESIGN AND PLAN

This open-label study will explore the impact of combination zonisamide and bupropion on the process of switching from combustible cigarettes (CC) to an e-cigarette.

Zonisamide is an FDA-approved medication with an anti-seizure indication, with daily doses usually ranging from 100 mg/day to 600 mg/day). It has multiple mechanisms of action, which include inhibiting activation of voltage-gated sodium channels at therapeutic levels. In addition, zonisamide also inhibits glutamate-mediated neurotransmission and enhances inhibitory GABA-ergic as well as serotonergic neurotransmission. It also enhances dopamine levels in the striatum, which in theory could help replace the desired effects of addictive drugs such as nicotine that also raise striatal dopamine. Topiramate, a drug sharing some actions with zonisamide, has been shown to facilitate smoking cessation and prevent post-cessation weight gain. Zonisamide has been shown to reduce ad libitum smoking as well as to relieve craving for cigarettes. It also has been shown to decrease anger, restlessness and impatience during smoking abstinence.

The zonisamide/bupropion combination has an additional rationale in that the potential side effects of each agent are offset by the other. For example, bupropion is associated with side effects of agitation and insomnia while zonisamide has sedative properties. Conversely, the side effects of zonisamide include sedation, which are expected to be partially offset by bupropion's stimulant actions. The combination of bupropion and zonisamide has been shown to be well tolerated in studies of weight loss produced by this drug combination.<sup>6</sup>

There is no therapeutic intent in that smokers' nicotine/tobacco dependence will not be treated; the goal is to switch from one form of nicotine/tobacco dependence (CC) to dependence on a different tobacco product (ecigarettes).

#### 1.2 BACKGROUND

According to the U.S. Surgeon General (2010 Report), the major smoking-related diseases, including cancer, heart and lung disease, have been linked to inhaling the combustion products of burning tobacco, rather than to nicotine per se. Therefore, less toxic forms of nicotine delivery, such as e-cigarettes, offer a potential avenue for harm reduction for smokers who cannot or do not wish to relinquish their nicotine dependence. A substantial fraction of smokers who use e-cigarettes continue to smoke combustible cigarettes ("dual use"), eroding the potential beneficial impact on disease risk. Therefore, it is important to examine strategies for enhancing complete switching to e-cigarettes from combustible cigarettes. We hypothesize that dual users find it most difficult to relinquish their favorite cigarettes, which surveys indicate are those smoked after meals. We hypothesize that a specific combination of FDA-approved medications shown to promote weight loss, consisting of bupropion and zonisamide, will reduce appetite, reduce the enjoyment of cigarettes after meals, and facilitate complete switching from combustible cigarettes to e-cigarettes. In addition to the hypothesized mechanism of reducing post-meal enjoyment of smoking, bupropion is an FDA-approved smoking cessation treatment (at 150 mg b.i.d.) that reduces craving for cigarettes as well as withdrawal symptoms of irritability, which could also facilitate complete switching. Bupropion and its metabolites block reuptake of dopamine and norepinephrine, which also have anti-depressant effects. 9

## 2 STUDY OBJECTIVES AND ENDPOINTS

#### 2.1 COMPLETE SWITCHING FROM CC TO HALO G6

The primary switching outcome will be smoking abstinence during weeks 8-11 post-quit date. This will be defined as self-report of no cigarette smoking (not even a puff), confirmed by an expired air CO reading of less than 5 ppm.

#### 2.2 Point Abstinence (From CC) at Six Months Post Switch

A secondary outcome will be 7-day point abstinence at 6 months post-switch, for participants who are smoking abstinent during weeks 8-11 post-quit, as defined above in Section 2.1. This will be assessed by self-report utilizing an automated SMS messaging system.

#### 2.3 Change in Rewarding Effects of Smoking Cigarettes

Secondary analyses will evaluate the hypothesis that enjoyment of smoking after meals is attenuated by zonisamide/bupropion treatment. The smoking satisfaction scale of the mCEQ-E will be compared between cigarettes smoked after meals versus all others smoked during the day, examining how this difference changes after zonisamide/bupropion usage. Additionally, the proportion of participants who report smoking after meals, while reporting not smoking at other times, will be compared between the first week and the weeks after zonisamide/bupropion usage.

# 3 INVESTIGATIONAL PLAN

#### 3.1 OVERALL STUDY DESIGN AND PLAN

This single-group, small-scale, open-label study (N= 25 to 50) will evaluate the impact of combination zonisamide and bupropion on the process of switching from combustible cigarettes (CC) to an e-cigarette. There will be a data collection period of at least five days to obtain baseline data on use of combustible cigarettes. Participants enrolled in the study will receive a G6 e-cigarette at V2 for *ad libitum* use. After the first week of e-cigarette use, (at V3) participants will be given zonisamide (100 mg/daily) and will begin extended-release bupropion dosing (150 mg each morning days 1-3, then 300 mg/daily) in addition to continued use of the G6. At each visit, participants will receive enough zonisamide, bupropion, and Halo G6 cartomizers to last until their next study visit. Halo G6 and combination zonisamide and bupropion use will continue until the participant returns for the End-of-Study visit (V7).



Figure 1 - Overall Study Design

The outcome of the combination zonisamide and bupropion on the process of switching from combustible cigarettes (CC) to an e-cigarette will be compared to the following benchmarks. Initial results will fall into one of the following three categories:

#### 3.1.1 Complete switching rate of 64%

If this study achieves at least a 64% (16/25) switching rate to Halo G6 for the first 25 smokers tested at V7, it will be viewed as having considerable promise, and will immediately be advanced to larger-scale (~N=200) randomized controlled clinical trials (RCTs) to provide a rigorous evaluation of its efficacy and effectiveness in helping smokers switch to e-cigarettes. Future trials will be submitted to the Institutional Review Board (IRB) as new protocols.

#### 3.1.2 Complete switching rate of 52% to 60%

If this study achieves switching to Halo G6 in 52%-60% (13/25 to 15/25) of the first 25 smokers tested at V7, then an additional sample of 25 smokers will be enrolled (total N=50) to obtain a more precise estimate of the switching rate. If, cumulatively, complete switching to G6 is achieved in at least 56% (28/50) at V7, the use of combination zonisamide and bupropion as an aid to switching will then be advanced to larger RCTs.

#### 3.1.3 Switching Thresholds Not Achieved

If either of the above switching rate thresholds is not met in the first 25-50 smokers tested, the use of combination zonisamide and bupropion as an aid to switching will be considered unpromising, and further participants will not be enrolled.

In choosing these thresholds, Monte Carlo simulations were conducted to determine the significance thresholds for both the N=25 and N=50 one-tailed binomial tests so that the overall false positive (Type I error) rate across all tests would be approximately 10%. Conversely, the overall false negative (Type II error) rate, whereby a promising procedure is discarded prematurely, would be approximately 20%. The diagram below depicts the stepwise evaluation algorithm.



#### 3.2 Study Procedures

At each session, expired air CO will be measured along with blood pressure, heart rate, respiratory rate and body weight. Participants will also complete questionnaires rating participantive effects of smoking and ecigarette use. Participants will be given enough cartomizers and study drugs to last until their next scheduled session, along with an extra 4 days' worth to allow for flexibility in case sessions need to be rescheduled. Ecigarette usage and study drug compliance will be tracked not only by self-reported number of occasions used, but also by cartomizer counts (used or unused) and returned study drugs.

#### 3.3 Point of Enrollment

Participants will be enrolled after all safety laboratory results have been received and reviewed by the medical staff (MD or PA). The Halo G6 and the cartomizers will be dispensed starting at V2, and at each subsequent visit until the End-Of-Study. Study drugs will be dispensed starting at V3, and at each subsequent visit until the End-Of-Study.

#### 3.4 STUDY AND SESSION DURATIONS

The total duration for a participant will be approximately 14-16 weeks. The Screening Session (Visit 1) will last approximately 2 ½ to 3 hours. The other study sessions will last approximately one hour.

# **4 PARTICIPANT INVOLVEMENT**

#### 4.1 SELECTION OF STUDY POPULATION

Healthy, cigarette smoking adults, age 21-65 years, with no restriction on gender, race and ethnicities, or social-economic status, who have smoked an average of at least 10 commercially available cigarettes per day for the last 12 months will be screened for enrollment in this study.

The study will screen and enroll at both Rose Research Center locations, located in Raleigh and Charlotte, North Carolina.

#### 4.1.1 Inclusion Criteria

Each participant must meet all the following inclusion criteria before enrollment:

#### **Inclusion Criteria**

- 1. Has signed the ICF and is able to read and understand the information provided in the ICF.
- 2. Is 21 to 65 years of age (inclusive) at screening.
- 3. Smokes at least 10 commercially available cigarettes per day (no brand restrictions), for the last 12 months.
- 4. Has an expired air CO reading of at least 10 ppm at screening.
- 5. Interested in switching to an electronic cigarette.
- 6. Willing and able to comply with the requirements of the study.
- 7. Owns a smart phone with text message and data capabilities compatible with necessary surveys.

#### 4.1.2 Exclusion Criteria

Potential participants who show or report indications of or self-report a diagnosis of conditions listed below may be excluded from the study. If the study physician (or designee) determines through the course of pre-screening, or a physical screen, medical history, physical findings, current medications, ECG, or laboratory findings suggests one of the conditions listed below, or findings reveal other information that may potentially jeopardize the participants' safe participation, then they may be excluded. For medical conditions that do not appear below,

the participant may be enrolled if the study physician (or designee) does not feel that the medical condition would jeopardize safe study participation or data validity.

Version 3.0 / 16 Feb 2021

#### **Exclusion Criteria**

- 1. Is unhealthy or cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason) as judged by the Investigator or designated medical staff based on all available assessments from the screening period (e.g., safety laboratory, vital signs, physical examination, ECG, concomitant medications and medical history).
- 2. PHQ-9 score greater than 9, or a score greater than 0 on item #9 ("Thoughts that you would be better off dead, or of hurting yourself in some way") at screening.
- 3. Planned use of an FDA-approved smoking cessation product during the study.
- 4. High blood pressure (systolic > 150 mmHg or diastolic >95 mmHg) at screening.
- 5. Body mass index (BMI) less than 15.0 kg/m<sup>2</sup> or greater than 40.0 kg/m<sup>2</sup>.
- 6. Coronary heart disease, structural cardiac disease (including, but not limited to valvular heart disease or cardiac murmurs), cardiac dysrhythmias, syncope, cardiac chest pain, or history of heart attack or heart failure.
- 7. Has received psychotherapy or behavioral treatments potentially impacting symptoms of depression, anxiety, or nicotine withdrawal within 30 days of screening, or during the study.
- 8. Taking antidepressants, psychoactive medications (e.g. antipsychotics, benzodiazepines, hypnotics) or medications that prolong QT<sub>c</sub>.
- 9. Use of any of these products in the past 30 days:
  - a. Illegal drugs (or if the urine drug screen is positive for cocaine, THC, amphetamines, methamphetamines, or opiates);
  - b. Experimental (investigational) drugs that are unknown to participant;
  - c. Chronic opiate use.
- 10. Use of smokeless tobacco (chewing tobacco, snuff), cigars (except for "Black & Mild" cigars or Cigarillos), pipes, hookah, e-cigarettes, nicotine replacement therapy or other smoking cessation treatments within 14 days of screening.
- 11. Pregnant or nursing (by self-report) or has a positive pregnancy test.
- 12. Enrollment requirements met.

#### 4.1.3 Women of Childbearing Potential

Pregnant or breastfeeding women will be excluded from the study. All females will undergo a serum pregnancy test at screening (Visit 1) and a urine pregnancy test at each subsequent visit. Heterosexually active females of childbearing potential (not post-menopausal) must agree to use medically acceptable contraceptives during the study. Medically acceptable contraceptives include: (1) surgical sterilization (such as a tubal ligation, hysterectomy, or Essure), (2) approved hormonal contraceptives (such as birth control pills, patches, implants or injections), (3) barrier methods (such as a condom or diaphragm) used with a spermicide, or (4) an intrauterine device (IUD). Contraceptive measures such as Plan B<sup>TM</sup>, sold for emergency use after unprotected sex, are not

acceptable methods for routine use. Female participants will be encouraged in the consent form to notify study staff if they believe a change in their pregnancy status has occurred during the trial.

Post-menopause is defined as the time after which a woman has experienced 12 consecutive months of amenorrhea (lack of menstruation).

#### 4.2 RECRUITMENT STRATEGIES

Participants will be selected through IRB approved generic recruitment advertisements which are specifically designed to recruit participants into the volunteer database for future smoking and tobacco use related research at the Rose Research Center. For this database, many of the participants have provided basic smoking history data along with demographic information, which will allow selection of potentially interested participants.

Participants who call in will be screened into the volunteer database, and if they pre-qualify, will be offered the option to prescreen for this protocol.

Participants will be contacted only with IRB approved appropriate materials and information submitted along with this protocol. These documents will include a brief description of the study and information on how to prescreen for participation. Participants will be contacted by phone, email and text message prompting interested participants to prescreen through an electronic screen form.

#### 4.2.1 Pre-Screening

Pre-screening will be completed prior to V1 for all participants. Participants will be provided with a set of IRB approved questions directly related to the inclusion and exclusion criteria. Based upon the outcome of these questions, potential participants may be scheduled for a screening visit (V1).

#### 4.3 Participant Retention in the Study

All candidates who schedule a screening visit (V1) will receive a series of email, text, and telephone reminders; participants are also permitted through these communications to confirm, cancel, or reschedule all their appointments.

#### 4.4 DISCONTINUATION OF PARTICIPANTS FROM STUDY

Discontinued participants will include both participants who withdraw from the study (participant's decision) or participants who are discontinued from the study (following Investigator's decision). A participant can only be discontinued from the study after enrollment. Participants that are not enrolled are considered screen failures.

Participants will be informed that they are free to withdraw from the study at any time. Participants should be questioned for the reason of premature withdrawal from the study, although they are not obliged to disclose it.

Participants discontinued from the study cannot re-enter the study.

#### 4.4.1 Participants will be discontinued from the study for any of the following reasons:

- Withdrawal of informed consent.
- Any adverse effect or condition that would jeopardize continued safe study participation.
- Pregnancy test is positive.

- Discontinuation is considered to be in the best interest for the participant or for other participants participating in the study, as judged by the Investigator or designee.
- 4.4.2 Participants may be discontinued from the study for any of the following reasons based on the judgment of the Investigator:

Version 3.0 / 16 Feb 2021

- No-show to appointments and unable to reschedule within the visit window.
- The misuse or abuse of study related equipment.
- Potential loss of the participant's data validity.
- Unwilling or unable to comply with study procedures.
- Enrollment discontinuation.

#### 4.5 LOST TO FOLLOW-UP

For participants lost to follow-up, a reasonable number of attempts to contact the participant (including written correspondence and/or phone calls) will be made and documented in the source documents. The date of the last contact (e.g. last visit, last phone call) will be recorded in the source document. When the PI (or designee) declares a participant is lost to follow-up, the lost to follow-up date will be recorded and will correspond to the date of the End of Study (EOS) of the participant.

## 4.6 VIOLATION OF INCLUSION/EXCLUSION CRITERIA

Participants who, after signing the ICF, do not meet the inclusion and exclusion criteria will not be enrolled in the study and will be considered screen failures. Re-screening for the study is not permitted.

#### 4.7 Participant Compensation

There will be a payment of \$25 for the Screening Session (V1) and \$75 at the completion of each study session V2 through V7. Participants will also receive an additional payment of \$5/day for responding to daily text messages during the 13-week product use period. If participants provide a CO reading at the six-month follow-up, they will receive an additional \$25.

If participants are asked by study staff to return to the center to complete or redo parts of the screening in situations of equipment malfunctions or other circumstances that are beyond the participants' control, participants may be reimbursed for mileage.

Participants who decide to withdraw from the study will be paid for the part of the study they have completed.

#### 4.8 Session and Response Windows

#### 4.8.1 V2 Session Window

Participants may attend V2 up to 30 days post Screening Session (V1).

#### 4.8.2 All other visit Windows

Participants may attend sessions up to four-calendar day's pre or post the scheduled visit.

#### 4.8.3 SMS Response Window

The SMS response window will be open until the next SMS message is sent.

# 5 HALO-G6 ELECTRONIC NICOTINE DELIVERY SYSTEM

#### 5.1 DESCRIPTION OF HALO G6

The Halo G6 is a breath-actuated, rechargeable e-cigarette that comes with prefilled e-liquid cartomizers. This ecigarette was chosen over other tank-based or pod-based e-cigarette models because of its similarity in shape and size to a cigarette. Because one of the goals is to provide habit substitution for smoking that zonisamide/bupropion cannot provide, this "cigalike" design is considered advantageous.

Version 3.0 / 16 Feb 2021

#### 5.2 DESCRIPTION OF E-LIQUID

Each G6 prefilled cartomizer contains a 50/50 blend nicotine salt with 35 mg nicotine strength. The 3.5% nicotine concentration was chosen over higher (e.g. 5%) concentrations to reduce the likelihood of nausea. The cartomizers come in packs of five. All Halo brand e-liquids undergo independent testing and they are manufactured by Nicopure labs. 10

This study will use "Tribeca" (tobacco) and "Menthol" flavored cartomizers, with participants matched to their preferred cigarette flavor. At Visit 2, participants will be allowed to use the device ad libitum for a maximum of 10 minutes. Research staff will inquire whether the participants are willing and able to use the Halo G6 during the study, to determine eligibility.

#### 5.3 PRODUCT USE TIMEFRAME

The maximum amount of time the G6 will be in use will be for 13 weeks, plus up to an additional four days (to allow for the scheduling window). Participants will be instructed on how to use the e-cigarette prior to dispensing.

#### 5.4 ACCOUNTABILITY AND COMPLIANCE

The G6 will be dispensed by the Investigator or designated study staff, as per study design. Participants will be dispensed cartomizers initially at 125% based on their daily smoking habits as reported at baseline (one per pack of cigarettes smoked per day). Participants may come into the office between visits to get additional supplies if needed. Each dispensation and collection of the product will be recorded.

#### Storage and Accountability

All products will be stored in a locked, limited-access area at the study site and kept at an ambient controlled room temperature, with excursions documented by RRC standard operating procedures. Halo products should not be exposed to extreme heat or cold.

#### 5.4.2 Compliance

Compliance will be ensured by strict distribution of the product and collection of devices (used and unused) which will be documented in appropriate logs.

# 6 ZONISAMIDE

#### 6.1 Description of Zonisamide

Zonisamide is currently marketed as an antiepileptic medication for treatment of partial seizures. While the main mechanism of action is believed to be related to its sodium and calcium channel blockade, the medication is suspected of exerting dose-dependent biphasic dopaminergic and serotonergic activity. As noted in Section 1.1, this medication has been shown to reduce ad libitum smoking and relieve craving from cigarettes. Zonisamide also has been shown to decrease anger, restlessness and impatience during smoking abstinence. The combination of bupropion and zonisamide has been studied as a treatment for weight loss in obese adults.

#### 6.2 Dosage

Dosing of zonisamide will remain unchanged for the duration of the 12-week dosing period unless changed per guidance below (section 6.3). Participants will take 100 mg (two 50 mg capsules) orally once a day.

#### 6.3 Dose Adjustment Procedures

Zonisamide will be dispensed in the form of a 50 mg capsules. Adjustments may be made to the timing of the dose (AM or PM) or the amount (1 or 2 capsules) depending on the somnolence/activation experienced by each individual participant. Initially, both bupropion and zonisamide will be taken in the morning. Should participants experience significant drowsiness, the medical providers (MD/PA) may change the dosing to nighttime (2 hours prior to bedtime) or decrease the dose to one 50 mg capsule per day. All dosing adjustments will be approved by the Medical Director for this study.

#### 6.4 ACCOUNTABILITY AND COMPLIANCE

#### 6.4.1 Dispensing Product

Zonisamide will be dispensed by the Investigator or designated study staff utilizing blister-pack technology to enhance compliance and accountability. Each dispense and collection of the product will be recorded during each laboratory visit (Visit 3 through Visit 6). All study-related drug will be collected at the End-Of-Study (Visit 7 or early termination).

Prior to dispensing, the site will ensure that the product packaging is labelled with the protocol number and unique participant identifiers, date it was dispensed, and the statements "For investigational use only" and "Keep out of reach of children".

#### 6.4.2 Storage and Accountability

Zonisamide will be stored in a climate-controlled secured-storage site with access limited to the authorized personnel only. Full accountability of the distributed products will be ensured by designated staff.

#### 6.4.3 Compliance

Compliance will be ensured by strict distribution of the product, daily SMS messages, and collection of unused products at each study session. This information will be documented in appropriate logs.

# 7 BUPROPION

#### 7.1 DESCRIPTION OF BUPROPION

Bupropion inhibits reuptake of both noradrenaline and dopamine. This medication has been approved as an antidepressant for over 20 years. The Food and Drug Administration approved the use of bupropion for smoking cessation in 1997. It is only one of two medications currently approved by the FDA for this purpose. The combination of bupropion and zonisamide has been studied as a treatment for weight loss in obese adults. The usual dose for bupropion for smoking cessation is 150 mg once a day for 3 days, followed by 300 mg once a day for 7 to 12 weeks. The maximum prescribed dose for bupropion is 450 mg a day, which is the maximum dose for treating major depressive disorder and attention deficit hyperactivity disorder for adults.

#### 7.2 Dosage

- 150 mg tablet orally once a day for 3 days.
- Two 150 mg tablets (300 mg) orally once a day for the remainder of study participation.

#### 7.3 Dose Adjustment Procedures

Bupropion will be dispensed in the form of a 150 mg extended release tablet, initially one tablet daily for 3 days, followed by 2 tablets daily until End of Study. Extended release tablets have a half-life that supports once daily dosing. Combining this medication with zonisamide will decrease the risk for side-effects, allowing for daily dosing, which will likely improve compliance. Adjustments will be made depending on the side-effects experienced by each individual participant. Initially, both bupropion and zonisamide will be taken in the morning. Should participants experience significant activation during the day, the medical providers (MD/PA) may either adjust the dose down to 150 mg daily or split the dose (150 mg taken twice daily which is normal dosing for smoking cessation). All dosing adjustments will be approved by the Medical Director for this study.

#### 7.4 ACCOUNTABILITY AND COMPLIANCE

#### 7.4.1 Dispensing Product

Bupropion will be dispensed by the Investigator or designated study staff utilizing blister-pack technology to enhance compliance and accountability. Each dispense and collection of the product will be recorded during each laboratory visit (Visit 3 through Visit 6). All study-related drugs will be collected at the End-Of-Study (Visit 7 or early termination).

Prior to dispensing, the site will ensure that the product packaging is labelled with the protocol number and unique participant identifiers, date it was dispensed, and the statements "For investigational use only" and "Keep out of reach of children".

#### 7.4.2 Storage and Accountability

Bupropion will be stored in ambient climate-controlled secured-storage site with access limited to the authorized personnel only. Full accountability of the distributed products will be ensured by designated staff.

#### 7.4.3 Compliance

Compliance will be ensured by strict distribution of the product, daily SMS messages, and collection of unused products at each study session. This information will be documented in appropriate logs.

Version 3.0 / 16 Feb 2021

### 8 STUDY PROCEDURES AND ACTIVITIES

Personnel performing study assessments must have appropriate and documented training. An overview of all study assessments is shown in the schedule of events (Section 7.5). Study personnel will adhere to standard operating procedures (SOPs) for all activities. Appropriate medical advice will be provided by qualified staff (licensed providers) to the participant in case of any medical findings requiring health care.

#### 8.1 Informed Consent and Guidance

Prior to any study assessments being performed, the participant will be asked to provide their written consent to participate in the study on an informed consent form (ICF). All assessments must start after the time of ICF signature by the participant for study participation.

Designated staff, under the supervision of the Principal Investigator, will obtain informed consent from each participant. The person obtaining consent provides the participants with a printed document that explains the procedures and risks. Designated staff will answer any questions. A signed copy of the informed consent form will be given to each participant. Participants are informed that they may withdraw from participation in the study at any time without penalty.

Because of the nature of this study and the number of questionnaires that participants are expected to complete, we do not recruit potential participants who do not read, are blind, or who do not understand English. We are not equipped to validate alternate versions of our questionnaires, most of which are not published. Questionnaires cannot be administered orally by a translator or by technicians to illiterate or blind participants because the data obtained would not be comparable to self-administered questionnaires.

#### 8.2 SAFETY LABORATORY AND OTHER ASSESSMENTS

An overview of all assessments is provided in the schedule of events.

Non-fasting blood samples and urine samples will be collected by qualified and trained site personnel. Participants will be in a seated or in a supine position during blood collection.

The maximal total volume of blood drawn for each participant will be around 30 mL for clinical chemistry, hematology, and serum pregnancy (for females).

Samples for clinical chemistry, hematology, and serum pregnancy test will be sent to LabCorp for analysis. Urinalysis will also be performed by LabCorp.

The results of the clinical chemistry, hematology and urine analysis safety panel will not routinely be given to participants to send or be sent to their physician to include in their medical record. However, if the participant's laboratory results are clinically relevant (including positive pregnancy tests), the research medical staff will send the participant a copy of the laboratory results. Participants who are accepted into the study but need medical

follow-up due to minor abnormalities in laboratory results (at any session) will also receive a copy of the laboratory results.

#### 8.2.1 Safety Laboratory

Safety laboratory includes clinical chemistry, hematology, and urinalysis and will be assessed at Visit 1.

#### 8.2.1.1 Clinical Chemistry

| Clinical Chemistry | |
|---|---|
| Sodium | Chloride |
| Potassium | Carbon dioxide |
| Blood urea nitrogen (BUN) | Creatinine |
| Glucose | Calcium |
| Total protein | Albumin |
| Bilirubin | Alkaline phosphatase (AP) |
| Aspartate aminotransferase (AST) | Alanine aminotransferase (ALT) |

#### 8.2.1.2 *Hematology*

| Hem | atology |
|---|---|
| Red blood cell (RBC) count | WBC count |
| Hemoglobin | Differential white blood cell (WBC) count |
| Hematocrit | Platelet count |
| Mean corpuscular volume (MCV) | Mean corpuscular hemoglobin concentration (MCHC) |
| Mean corpuscular hemoglobin (MCH) | |

#### 8.2.2 Urine Samples

Urine samples will be collected for the urine drug screen (at screening session), urine pregnancy test (at all sessions except screening), and safety urinalysis (at screening session). The urine drug screen and pregnancy tests will be performed by study personnel at the study site. The urine sample collected for urinalysis will be sent to LabCorp for testing.

In case of any positive pregnancy test, the Investigator or designee will inform the participant about the risks associated with smoking during pregnancy.

In the event of a positive urine drug test for cocaine, THC, opiates, amphetamines, or methamphetamines at the screening visit (V1), participants are notified that they have been excluded from study participation because of a positive drug test.

| Urinalysis |
|-----------------------|
| рН |
| Red blood cell traces |
| Bilirubin |
| Protein |
| Glucose |
| Specific gravity |
| Nitrite |
| WBC Esterase |

Table 1 - Urinalysis Assessments

| Drug Screening |
|-----------------|
| Amphetamine |
| Cocaine |
| THC |
| Methamphetamine |
| Opiates |

Table 2 - Drug Screening

#### 8.2.3 Serum Pregnancy Test

Serum pregnancy test will be performed during the screening visit for all females.

| Serum Pregnancy Test |
|-------------------------------------------------|
| Quantitative human chorionic gonadotropin (HCG) |
| test |

#### 8.2.4 Urine Pregnancy Test

The urine pregnancy test will be performed by study personnel on site for all females at each visit (except screening).

#### 8.2.5 Electrocardiogram (ECG)

ECG recording will be performed as per the site's standard operating procedures. A standard 12-lead ECG will be recorded after the participant has rested for at least 5 minutes in a supine position.

The following parameters will be documented: heart rate, PR interval, QRS interval, QT interval, and QTc interval. Every ECG will be assessed as normal, abnormal – not clinically significant, or abnormal – clinically significant.

ECG print-outs will be interpreted by a qualified physician or licensed medical provider. Any print-outs of ECGs on thermo-sensitive paper must be photocopied and stapled together for inclusion in the source documents and signed by the Investigator or designee.

#### 8.2.6 Vital Signs

Vital signs (systolic and diastolic blood pressure, pulse rate, temperature and respiratory rate), will be measured in sitting position after the participant has rested for at least 5 minutes. After two minutes of standing, a second blood pressure reading (systolic and diastolic) and pulse rate will be obtained at the screening visit (V1).

#### 8.2.7 Physical Examination

A complete physical examination, including auscultation and palpation will be performed. A complete physical examination will include review of general appearance, hair and skin, head, eyes, ears, nose and throat, neck, chest, abdomen, dentition, cardiovascular, musculoskeletal and neurological systems. The physical examination is to be conducted by a designated fully trained representative.

Appropriate medical recommendations will be provided to the participant if any medical findings requiring health care are identified.

#### 8.2.8 Expired Air CO Breath Test

Carbon Monoxide (CO) in participant's exhaled breath (expressed as ppm) will be measured using a Vitalograph CO Monitor. Participants must have an expired air CO reading at V1 of at least 10 ppm for inclusion into this study. This test will be repeated at each of the sessions.

#### 8.2.9 Medical History and Concomitant Disease

Relevant medical history and concomitant disease will be documented at the screening visit (V1). Medical history is defined as any condition that started and ended prior to screening. A concomitant disease is defined as any condition that started prior to screening and is still ongoing at V1 (this may also include findings detected during the screening visit (V1)).

#### 8.2.10 Prior and Concomitant Medication

All medication taken 30 days prior to the screening visit (V1) and during the study will be documented. Medications which are stopped before the screening visit (V1) will be considered as prior medication. Medications which are started prior to the screening visit (V1) and which are still being taken by the participant during the study, as well as medications that are initiated after the screening visit (V1) will be considered as concomitant medications. This applies to both prescription and over-the-counter products (e.g., vitamins).

Records of prior and concomitant medications taken include the drug name (preferably both generic and trade name), route of administration, dose/unit, frequency of use, indication, the start and, if applicable, the stop date. Any therapy changes (including changes of regimen) during the study will be documented.

#### 8.2.11 Body Height and Body Weight

Body weight will be measured at each visit. Height and weight will be measured at screening, and body mass index (BMI) will be calculated.

#### 8.2.12 Demographics

Sex, date of birth, race and ethnicity will be recorded for each participant according to Section 8.5.

#### 8.2.13 AE/SAE Reporting

AEs/SAEs will be assessed using questionnaires and interviews at the indicated time points and spontaneous reporting from the time of ICF signature until the EOS for the participant (see Section 8.5).

#### 8.2.14 Questionnaires

The questionnaires will be administered to the participants using paper questionnaires and/or an electronic data collection system. The questionnaires will be asked according to Section 8.5.

#### 8.2.14.1 PHQ-9 -- The Patient Health Questionnaire

The Patient Health Questionnaire PHQ-9 for Depression will be used to screen for current (within 2 weeks) depression. Potential participants who score >9 (or who score >0 on item #9 ("Thoughts that you would be better off dead, or of hurting yourself in some way")) will be excluded from study participation, and, at the discretion of the study physician/physician assistants, referred to appropriate psychiatric treatment. Participants will respond to this questionnaire at all visits. This questionnaire will be administered at every visit, including the screening visit (V1 through V7).

# 8.2.14.2 Modified Cigarette Evaluation Questionnaire-Extended (mCEQ-E) and Modified Electronic Cigarette Evaluation Questionnaire-Extended (mECEQ-E)

The Cigarette Evaluation Questionnaire was initially developed in the PI's laboratory and used in numerous studies to assess the effects of pharmacological treatments on the rewarding effects of cigarette smoking. The mCEQ-E will be utilized to assess the degree to which participants experience the reinforcing of smoking, providing five subscale scores: smoking satisfaction (satisfying, tastes good, enjoy smoking), psychological rewards (calms down, more awake, less irritable, helps concentrate, reduces hunger), aversion (dizziness, nauseated), enjoyment of respiratory tract sensations (single-item assessment), craving reduction (single-item assessment). Participants will be asked to assess the 12 items of the questionnaire on a 7-point scale, ranging from "not at all" to "extremely". These 12 items will be asked for the "first cigarette smoked", "cigarette immediately after a meal", and "all other cigarettes." The e-cigarette version of this questionnaire (mECEQ-E) will also be used.

#### 8.2.14.3 Shiffman-Jarvik Withdrawal Scale

The Shiffman-Jarvik Withdrawal Scale is used to measure withdrawal symptoms and a participant's desire to smoke. This scale consists of five subscales: craving, psychological symptoms, physical symptoms, sedation, and appetite.<sup>13</sup>

#### 8.2.14.4 Reasons to Smoke

The Reasons to Smoke questionnaire (Appendix 17) is used to determine the most important reasons to smoke for each participant.

#### 8.2.14.5 FTND -- The Fagerström Test for Nicotine Dependence

The Fagerström Test for Nicotine Dependence is a six-item questionnaire developed by Karl-Olov Fagerström and is used to determine someone's level of nicotine dependence. The scores obtained on the test allow the classification of nicotine dependence in three different levels: mild (0-3 points), moderate (4-6 points), and severe (7 -10 points).

#### 8.2.14.6 ABOUT – Assessment of Behavioral Outcomes

The ABOUT is a self-report instrument that measures dependence in a directly comparable way across different tobacco- and nicotine-containing products.

#### 8.2.14.7 Prior and Concomitant Medication

At each visit, participants will report any changes in medication use, including the use of supplements, vitamins, over-the-counter medications, and prescription medications.

#### 8.2.14.8 Smoking History Questionnaire

The Smoking History is a questionnaire designed to help assess the participant's current and past smoking habits. This questionnaire will be administered at screening (V1) and will include questions about the number of years participants have smoked combustible cigarettes (CC), the number of CCs per day smoked over the last 12 months, brand of CCs, use of other tobacco products and use of nicotine replacement therapy or other smoking cessation treatments. This questionnaire will also be used to check eligibility criteria.

#### 8.2.14.9 Registration Form

This form is an internal questionnaire designed to collect demographic information about participants. It will be administered at screening (V1).

#### 8.2.14.10 Medical History Form

The Medical History form is an internal questionnaire designed to help assess the participant's current health and any health history. This questionnaire also includes questions about all medications (include prescription medications, other-the-counter medications or supplements) taken in the past 30 days. It is designed to help assess the participant's current health and health history and is used to help determine eligibility. This form is administered at the initial screening visit (V1).

Version 3.0 / 16 Feb 2021

#### 8.2.14.11 Review of Systems

The Review of Systems is an internal questionnaire administered at screening (V1) to help assess the participant's current health and health history by asking about the presence of a list of symptoms.

#### 8.2.14.12 *Employment History*

The Employment History is an internal questionnaire designed to collect information about a participants' social economic status. Participants will be presented this questionnaire after enrollment, at the second visit (V2).

#### 8.2.14.13 *Medication Compliance*

Participants will be queried via SMS text messages whether they have been compliant with taking the study specific medications. These messages will commence after the second visit and continue through the End of Study.

#### 8.2.14.14 *Smoking Status*

SMS text messages will be sent to participants starting after enrollment, through the End of Study, to ascertain the participants smoking status.

#### 8.3 5-Day Smoking Baseline Collection

After verification of eligibility (approximately two days after screening), participants will commence a five-day smoking baseline data collection. Participants will be called and given instructions on the use of the SMS system which will administer questions about smoking status in order to collect baseline data prior to start of the Halo and the study drugs.

#### 8.4 6-Month Follow Up

Participants who complete the study will be contacted six months after the switch day utilizing an automated SMS messaging system, to ascertain their current smoking status and use of e-cigarettes. If a participant selfreports current abstinence from smoking they will be asked to return to the office for collection of an expired air CO for verification.

# 8.5 SCHEDULE OF EVENTS

| | Visit Assessments and Procedures Screening Session Cig Data Collection | | V2 | Product<br>Use Period<br>13 Weeks<br>PM SMS | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Informed Consent and Guidance | • | | | | | | | | |
| | Inclusion/Exclusion Criteria | • | | | | | | | | |
| | Enrollment/Randomization | | | • | | | | | | |
| | Prior and Concomitant Medication | • | | • | • | • | • | • | • | |
| | Smoking History Questionnaire | • | | | | | | | | |
| | Registration Form | • | | | | | | | | |
| | Employment History | | | • | | | | | | |
| | Medical History/Review of Systems | • | | | | | | | | |
| | Payment Verification Form | • | | • | • | • | • | • | • | |
| ires | Reasons to Smoke | | | • | | | | | •* | |
| Questionnaires | Modified Cigarette Evaluation Questionnaire Extended (mCEQE) | | | • | • | ٠ | • | • | • | |
| stio | $Modified\ e\hbox{-Cigarette Evaluation Question naire Extended (meCEQE)}$ | | | | • | ٠ | • | • | • | |
| Jue | The Fagerström Test for Nicotine Dependence (FTND) | | | • | • | | | | • | |
| | Shiffman-Jarvik Withdrawal Scale | | | ٠ | • | ٠ | ٠ | • | ٠ | |
| | Assessment of Behavioral OUTcomes (ABOUT) | | | ٠ | • | | | | • | |
| | Patient Health Questionnaire (PHQ-9) | • | | • | • | ٠ | • | • | • | |
| | e-Cigarette Usage and Smoking Status (via daily SMS text) | | • | | | | | | | • |
| | Medication Adherence (via daily SMS text) | | | | | | | | | • |
| | Safety Laboratories | • | | | | | | | | |
| | Serum Pregnancy Test (Females) | • | | | | | | | | |
| | Urine Pregnancy Test (Females) | | | • | • | ٠ | • | • | • | |
| | Urine Drug Screen | • | | | | | | | | |
| | CO Breath Test | • | | ٠ | • | ٠ | ٠ | • | • | |
| | ECG | • | | | | | | | | |
| | Blood Pressure | • | | • | • | ٠ | • | • | • | |
| S | Heart rate | • | | • | • | • | • | • | • | |
| Vitals | Temperature | • | | | | | | | | |
| _ | Respiratory rate | • | | • | • | • | • | • | • | |
| | Weight | • | | • | • | • | • | • | • | |
| | Height | • | | | | | | | | |
| | Physical Examination | • | | •# | •# | •# | •# | •# | •# | |
| Halo Assessment and Questionnaire Collect Used/Unused Halo products Dispense Halo products | | | | • | | | | | | |
| | | | | | • | ٠ | • | • | • | |
| | | | | • | • | ٠ | • | • | | |
| Collect Used/Unused Blister Packs | | | | | | ٠ | • | • | • | |
| Dispense Study Drugs in Blister Packs | | | | | • | • | • | • | | |

<sup>#</sup> Targeted examination as needed

<sup>\*</sup> Based on current product use

#### 8.6 SMS Messaging

- 8.6.1 Daily SMS Message (after screening, prior to V2) Participants will receive a text with a link to a survey to access the following:
  - Have you smoked any combustible cigarettes today?
    - o If yes, how many cigarettes did you smoke?
    - What was your favorite cigarette of the day?
       1-First one, 2-One immediately after a meal, 3-Any other cigarette
- 8.6.2 Daily SMS Message (From Visit 2) -- Participants will receive a text with a link to a survey to assess the following:
  - Have you smoked any combustible cigarettes today?
    - o If yes, how many cigarettes did you smoke?
    - Which cigarette did you smoke today? (If only 1 cigarette is reported)
       1-First one of the day, 2-One immediately after a meal, 3-Any other cigarette
    - What was your favorite cigarette of the day? (Of more than 1 cigarette is reported)
       1-First one, 2-One immediately after a meal, 3-Any other cigarette
  - Have you used your e-cigarette today?
    - o If yes, how many times did you use your e-cigarette today?
  - Did you take your study drugs this morning? (After Visit 3)
- 8.6.3 6-Month follow up SMS Message -- Participants will receive a text with a link to a survey to assess the following:
  - Have you smoked a combustible cigarette since your last visit?
    - o If yes, are you still smoking combustible cigarettes right now?
    - o How many combustible cigarettes do you smoke per day on average?
  - Have you used an e-cigarette since your last visit?
    - o If yes, are you still using an e-cigarette?
    - O How often do you use an e-cigarette?
  - Have you used any other nicotine containing products (other than e-cigarettes) since you last visit?

# 9 RISK / BENEFIT INFORMATION

#### 9.1 POTENTIAL RISKS

Continuing to smoke carries significant health risks; however, the participants in the studies will have expressed an interest in switching from smoking combustible cigarettes to using an electronic cigarette during the brief study duration, and hence will not be exposed to significant additional risks.

#### 9.1.1 Zonisamide

The most common adverse effects of zonisamide include somnolence, dizziness, nausea, heartburn, constipation, weight loss, changes in taste, dry mouth, drowsiness and headache. In prior clinical trials of zonisamide, discontinuation rates varied between 4% to 24% due to adverse effects (these studies

administered daily doses of 300 to 500 mg).<sup>14</sup> This study will evaluate zonisamide at a maximum dose of 100 mg daily.

#### 9.1.2 Bupropion

Common adverse effects of bupropion (occurring greater than 5% more than placebo) include headache, dry mouth, nausea, insomnia, constipation, and dizziness. These adverse effects were observed for doses ranging from 300 mg to 400 mg daily. Adverse events leading to discontinuation in clinical trials occurred at a relatively low rate, with 7% drop-out for all doses, 9% drop-out at the 300 mg dose, and 11% drop-out for the 400 mg dose. This study will utilize bupropion at a maximum dose of 300 mg daily. <sup>15</sup>

#### 9.1.3 Use of Halo G6

The common risks associated with e-cigarette use include coughing, dry mouth, throat irritation, sore throat and shortness-of-breath.

#### 9.1.4 Tobacco Withdrawal

To the extent that nicotine or other tobacco smoke constituent intake is reduced or eliminated, participants may experience tobacco withdrawal symptoms, including craving, difficulty concentrating, mood disturbance and increased appetite/weight gain.

#### 9.1.5 Nicotine Toxicity

The e-cigarette may deliver less of various tobacco smoke constituents than participants' usual brands of cigarettes, and in some cases, may deliver more nicotine. However, participants control their nicotine intake and many studies have shown that smokers effectively limit their nicotine intake from cigarettes to avoid symptoms of nicotine toxicity (e.g., nausea, vomiting, sweating, headache, dizziness, jittery, palpitations, or in the case of extreme cases of nicotine overdose, convulsions, respiratory paralysis and death).

#### 9.1.6 Blood Draw

The risks associated with venipuncture are minimal and include momentary discomfort and/or bruising. Infection, excess bleeding, clotting, and fainting are also possible, although unlikely.

#### 9.2 Protection Against Risks

The risks to which participants will be exposed are comparatively minor, because it is unlikely when using the e-cigarette that they will be exposed to higher levels of toxicants than when smoking their cigarettes. Smokers are very experienced in regulating their nicotine intake to avoid excessive amounts. Additionally, participants will be screened medically and monitored throughout the study.

Study participants will receive detailed instructions on the use of the tobacco products distributed to them, in order to minimize the possibility of misuse. Participants will be instructed to keep all nicotine/tobacco products away from children and pets.

Participants will be instructed to report any side effects to study staff, who will communicate these reports to the medical staff. The most appropriate course of action will be determined, which may include options for termination of exposure to study-related clinical materials (e.g., e-cigarettes), options for dose modifications to study drugs, or complete termination of study drugs. Participants will,

however, be reminded that they have the option to withdraw from the study at any time. Participants will also be given a 24-hour emergency contact number in the event that side effects or adverse events occur between sessions.

# 10 QUALITY CONTROL AND QUALITY ASSURANCE

#### **10.1** Training of Staff

The Investigator or designee will ensure that appropriate training relevant to the study is provided to all staff involved in the study, and that any new information relevant to the performance of this study is forwarded in a timely manner to the staff.

#### **10.2** AUDITS AND INSPECTIONS

Good Clinical Practice regulations require independent inspections of clinical program activities. Such inspections may be performed at any time before, during, and after the study.

Authorized representatives of the Sponsor, regulatory agencies and/or an IRB may perform audits or inspections, including source data verification. The purpose of an audit or inspection is to systematically and independently examine all study-related activities and documents to determine whether these activities were conducted, and data were recorded, analyzed and accurately reported, according to the protocol, ICH/GCP guidelines and any applicable regulatory requirements. The Investigator or designee will contact the Sponsor immediately if contacted by a regulatory agency about an inspection at their site.

The Investigator and study staff are responsible for maintaining a comprehensive and accurate filing system of all study-related documentation that will be suitable for inspection at any time by the Sponsor, its authorized representative, and other regulatory agencies.

# 11 REPORTING OF ADVERSE EVENTS

#### 11.1 DEFINITIONS

#### 11.1.1 Adverse Event

An Adverse Event (AE) is defined as any untoward medical occurrence that may present during participation in the study and which may or may not have a causal relationship with study procedures and/or products tested in this study. An adverse event (AE) can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the study procedures and/or products.

Any increase in the severity and/or the frequency of a concomitant disease is considered an AE.

#### 11.1.2 Serious Adverse Event

A Serious Adverse Event is any adverse event that:

- results in death;
- is life-threatening;
- results in inpatient hospitalization or prolongation of existing hospitalization;
- results in persistent or significant disability / incapacity;
- results in a congenital anomaly / birth defect;
- requires immediate medical or surgical intervention.

Important medical events that may not result in death, be life threatening, or require hospitalization may be considered an SAE, when, based on appropriate medical judgment, the event may jeopardize the participant, or the participant may require medical or surgical intervention to prevent one of the outcomes listed in the above definitions.

The term "life-threatening" in the definition of "serious" refers to an event in which the participant was at risk of death at the time of the event; it does not refer to an event, which hypothetically might have caused death if it were more severe.

Any pre-planned hospitalizations that are known at the time of signing the ICF will not be recorded as an SAE; however, they will be recorded as AE only. Any AE that occurs during this pre-planned hospitalization will be considered according to the above definitions.

#### 11.2 COLLECTION OF SAFETY EVENTS FROM PARTICIPANTS

Information recorded when collecting AEs will include: thorough description of the AE, seriousness assessment, start and stop dates (if known), circumstances leading up to the event, clinical elements such as clinical course, specific vital signs and test results that may explain the pathophysiology of the event, as well as alternative explanations to its occurrence, the action taken with the investigation product/procedures due to the AE, the participant's disposition in the study after the occurrence of the AE and the final outcome of the AE (if known).

Any exacerbation/worsening or increased frequency of an AE or pre-existing condition shall be evaluated and recorded.

AEs should be collected using interviews with the participant.

Whenever a medically meaningful diagnosis is available to comprise a set of reported signs and/or symptoms, it should be preferentially provided as the AE or SAE term, rather than the individual signs and/or symptoms. Otherwise, each one of those signs and/or symptoms should be reported separately as event terms.

#### 11.2.1 Period of Collection

All existing health conditions identified during the Screening Period will be recorded as concomitant disease and the participant's eligibility will be reviewed. Any AEs which occur during the screening session will be captured by the study site staff and assessed by the Investigator or designee in order to establish relationship or relatedness in respect to study procedures.

Any new, clinically relevant, abnormal finding detected during the study or worsening of a pre-existing condition/concomitant disease will be documented as an AE or an SAE.

All ongoing AEs at the End of Study participation will be followed-up by the Investigator or designee until they have improved, resolved, stabilized (i.e., no worsening of condition), or until an acceptable explanation has been found. The Investigator or designee will refer the participant to their Primary Care Provider for follow up of those AE when appropriate.

#### 11.3 Assessment of Adverse Events

#### 11.3.1 Intensity of Adverse Events

For each AE/SAE, the intensity will be graded on a 3-point intensity scale:

- Mild: The AE is easily tolerated and does not interfere with daily activity.
- Moderate: The AE interferes with daily activity, but the participant is still able to function.
- Severe: The AE is incapacitating and requires medical intervention.

#### 11.3.2 Relationship to Study Procedures

In general, all AEs and SAEs will be assessed by the Investigator or designee as either 'related' or 'not related'.

- Not related: The temporal relationship of the clinical event to study procedures and/or the study medication makes a causal relationship unlikely, or, concomitant medication, therapeutic interventions, or underlying conditions provide a sufficient explanation for the observed event.
- Related: The temporal relationship of the clinical event to study procedures and/or the study
  medication makes a causal relationship possible, and concomitant medication, therapeutic
  interventions, or underlying conditions do not provide a sufficient explanation for the
  observed event.

#### 11.3.3 Expectedness Assessment

All AEs and SAEs will be assessed by the Investigator or designee as either 'expected' or 'unexpected'. The determination of expectedness for an event is based upon the judgement of the Investigator (or designee). An 'unexpected' AE/SAE occurs with a nature/severity/incidence that has not previously been observed or reported and is inconsistent with the known risk information described in literature and/or as listed in this protocol.

#### 11.4 FOLLOW-UP OF NON-SERIOUS AND SERIOUS ADVERSE EVENTS

All ongoing Non-Serious AEs at the End of Study participation will be followed-up by the Investigator or designee until they have improved, resolved, stabilized (i.e., no worsening of condition), or until an acceptable explanation has been found. The Investigator or designee will refer the participant to their Primary Care Provider for follow up of those AE when appropriate.

Serious AEs will be followed up by the Investigator or designee, despite their continuation after the End of Study, until their resolution, stabilization (i.e., no worsening of the condition), or an acceptable explanation has been found (e.g. a chronic condition).

#### 11.5 Reporting of Safety Events to IRB

The Principal Investigator will report all serious adverse events relating to the study in an expedited manner to the Institutional Review Board (IRB) office in accordance with the Center's standard operating procedures and GCP reporting guidelines.

#### 11.6 REPORTING OF SAFETY EVENTS TO FDA

The Principal Investigator will report any suspected adverse reaction to study treatment that is both serious and unexpected to the FDA following established Safety Reporting guidelines.

#### 11.7 REPORTING AND FOLLOW-UP OF PREGNANCIES

All participants who are determined to be pregnant after enrollment will be discontinued from the study. Advice on the risk of smoking and smoking cessation will be provided by the study doctor (or qualified staff) and participants will be referred to the respective health care facility/health care provider for further support.

The Investigator is responsible for informing the IRB of any pregnancy that occurs during the study according to local regulations.

#### 11.8 Adverse Event Leading to Discontinuation

If a participant is discontinued from the study because of an AE, the Investigator or designee will follow up until the AE(s) has/have been resolved, stabilized (i.e., no worsening of condition), or until an acceptable explanation has been found.

#### 12 DATA MANAGEMENT

#### 12.1 DATA COLLECTION PROCEDURES

The results from the clinical assessments will be recorded in the source data file by the Investigator or their authorized designee and then captured in the case report forms (CRFs), unless otherwise specified in the final protocol. Trained study personnel will be responsible for capturing the data from the observations, tests, and assessments specified in the protocol and in the source documents. Study personnel will transfer the data to the CRFs.

The Investigator has ultimate responsibility for the collection and reporting of all data related to the clinical study and ensuring that the data are accurate, authentic/original, legible, timely (contemporaneous), enduring, and available when required. Any corrections made to source documents must be clearly recorded, without obscuring the original values and be accompanied by the date of change, reason for change, and identification of the person making the change. CRF data will be verified against the source documents at the study site by appropriate staff. Instances of missing or unclear data will be discussed with the Investigator for resolution.

#### 12.2 Protocol Deviations / Noncompliance

Protocol deviations are defined as deviations from the study procedures as defined in this document, whether intentional or unintentional that may affect the participant's rights, safety, or well-being and/or the completeness, accuracy and reliability of the data.

Noncompliance that meets the above definition must be reported to the IRB within 10 days of becoming aware of the noncompliance.

#### 12.3 DATA CAPTURE

All data are collected from participants using paper documents or an electronic data capture system. All applicable data, as specified in the protocol, will be transferred to the database or applicable Case Report Forms.

#### 12.3.1 Salesforce.com

Data will be collected for recruitment and screening purposes as stated within an Advarra IRB generic recruitment protocol. Unrelated to that protocol, pre-screening questionnaires will be attached to potential participant's records on whether they qualify or are disqualified for this study. Questionnaires utilized for this study will be permanently attached to that potential volunteer's record unless that information is requested to be removed by the participant.

#### 12.3.2 Survey Monkey

Survey Monkey uses some of the most advanced technology for Internet security that is commercially available today. This Security Statement is aimed at being transparent about our security infrastructure and practices, to help reassure that data is appropriately protected. Visit Survey Monkey privacy policy for more information on data handling.

All Survey Monkey information systems and infrastructure are hosted in world-class data centers. These data centers include all the necessary physical security controls you would expect in a data center these days (e.g., 24×7 monitoring, cameras, visitor logs, entry requirements). SurveyMonkey has dedicated cages to separate our equipment from other tenants. In addition, these data centers are SOC 2 accredited.

#### 12.3.3 Short Message Service (SMS) Messaging

SMS Messaging will be utilized for the delivery of a hyperlink to a mobile device to collect study data. This data will be collected utilizing an electronic survey. The service utilized for these messages is textit.in.

#### 12.3.4 Medrio

All smoking behavioral and self-report measures will be captured initially using Medrio. Medrio is an electronic data collection system that records and performs analysis and reporting of data. Participant data will be kept within Medrio's secure servers and may only be transmitted through a secure (SSL) download to our local server. Medrio's servers are protected by high-end firewall systems, with vulnerability scans performed regularly. All services have quick failover points with redundant hardware, and complete encrypted backups are performed regularly. Medrio uses Transport Layer Security (TLS) encryption (SSL or HTTPS) for all transmitted internet data. All information collected within Medrio is compliant with 21 CFR 11 requirements.

#### 12.4 DATA HANDLING

Data of all participants enrolled including screening failures and AE/SAEs during the study (from the time of informed consent to the end of the study of the participant) will be captured in the source documents.

# 13 PLANNED STATISTICAL METHODS

All data measures (e.g., withdrawal symptoms questionnaires, smoking history, smoking diaries, etc.) are captured initially using paper or an electronic data capture system. Verified data files will be analyzed using Statview or SAS (Statview, SAS Institute, Cary NC). Data will be inspected for outliers and if sufficiently extreme (Chauvenet's criterion, after verifying normality of distributions) will be censored from the data analysis.

#### 13.1 OUTCOMES

#### 13.1.1 Switching Outcome

Complete switching from combustible cigarette use at each time point will be defined by a self-report of no cigarette smoking (not even a puff) since the prior session, confirmed by an expired air CO reading of less than 5 ppm. The primary switching outcome will be smoking abstinence during weeks 8-11 post-switching date. An intent-to-treat approach will be taken in which any participants lost to follow-up after the point of randomization, or who have smoked during weeks 8-11 will be counted as having not completely switched to e-cigarette use. A secondary outcome will be 7-day point abstinence at 6 months post-switch. The main goal of the 6-month follow-up is to assess the persistence of switching to e-cigarettes. The main hypothesis to be evaluated in this pilot study is that the rate of complete switching to e-cigarette use will be greater than the historical benchmark of 45% smoking abstinence expected with varenicline when it is used in smoking cessation treatment.

#### 13.1.2 Change in Rewarding Effects

Change in reported rewarding effects of smoking for cigarettes smoked in the morning, after meals and at other times during the day will be compared.

#### 13.2 Interim Analysis

An interim analysis will be conducted after results are collected from the first 25 participants, in order to determine whether the trial will stop, or an additional 25 participants will be enrolled, as described above.

# 14 ETHICS AND REGULATIONS

#### 14.1 IRB APPROVAL

The protocol, informed consent document and relevant supporting information must be submitted to the IRB for review and must be approved before the study is initiated. In addition, any participant recruitment materials must be approved by the IRB prior to being used.

Any change to the protocol must be submitted to the IRB for review and approval before implementation. A protocol change intended to eliminate an apparent immediate hazard to participants may be implemented immediately provided the reviewing IRB are notified within 10 working days.

#### 14.2 Investigational New Drug Application

An Investigational New Drug (IND) application is not required for use of zonisamide or bupropion in this study. This study is not intended to support a new indication, support a change in labeling, support a change in advertising, nor does it involve a change in dosage level or route of administration.

An Investigational New Drug (IND) application is not required for use of Halo G6 in this study because the G6 is not intended for use as a smoking cessation aid.

#### 14.3 Investigational Tobacco Product Application

An Investigational Tobacco Product (ITP) application is not required for use of the Halo G6 in this study. The device and the cartomizers were marketed prior to August 8, 2016 and are not being modified for the investigation.

#### **14.4 GCP** AND REGULATORY REQUIREMENTS

This study will be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki and that are consistent with Good Clinical Practice and applicable regulatory requirements. The study must be conducted in accordance with the regulations of the United States Food and Drug Administration (FDA) as described in 21 CFR 50 and 56, applicable laws and the IRB requirements.

#### 14.5 Participant Information and Consent

It is the responsibility of the investigator to provide each participant with full and adequate verbal and written information using the IRB-approved informed consent form (ICF), including the objective and procedures of the study and the possible risks involved before inclusion in the study. Informed consent must be obtained prior to performing any study-related procedures.

The signed and personally dated original and completed ICF(s) must be kept by the Investigator and filed in the Investigator study file at the site or with the participant's files and a copy must be given to the participant. The participant will be informed that if they discontinue from the study, the data collected until the point of discontinuation will be maintained as part of the study data and the samples collected prior to discontinuation will be analyzed, unless they refuse in writing.

#### 14.6 AMENDMENT TO INFORMED CONSENT FORM

If a protocol amendment is required, an amendment may be required to the ICF. If revision of the ICF is necessary, the Investigator or designee will ensure that the documents have been reviewed and approved by the IRB before participants are informed and sign the amended ICF (including date and time).

# 15 Administrative Considerations

#### 15.1 Participant Confidentiality

All information obtained during the conduct of the study with respect to the participants' state of health will be regarded as confidential. A statement to this effect will be written in the information provided to the participant. An agreement to disclose any such information will be obtained from the participant in writing and signed by the participant, in compliance with all local and national data protection and privacy legislation.

Study records that identify participants will be kept confidential as required by law. Except when required by law, participants will not be identified by name, social security number, address, telephone number, or any other direct personal identifier in study records disclosed outside of Rose Research Center. For records disclosed outside of Rose Research Center, participants will be assigned a unique code number. The key to the code will be kept separate from the locked file where the study records are stored.

#### 15.2 RECORD RETENTION

All records of data, in any form, will be maintained by Rose Research Center as required by ICH/GCPs. Essential documents will be retained for at least 15 years after completion of the study.

Appropriate measures will be taken to prevent accidental or premature destruction of these documents.

# 16 REFERENCES

- 1. Kadian R, Kumar A. Zonisamide. In: *StatPearls*. Treasure Island (FL): StatPearls Publishing; 2020. http://www.ncbi.nlm.nih.gov/books/NBK507903/. Accessed March 2, 2020.
- 2. Biton V. Clinical pharmacology and mechanism of action of zonisamide. *Clin Neuropharmacol*. 2007;30(4):230-240. doi:10.1097/wnf.0b013e3180413d7d
- 3. Leppik IE. Zonisamide: chemistry, mechanism of action, and pharmacokinetics. *Seizure*. 2004;13 Suppl 1:S5-9; discussion S10. doi:10.1016/j.seizure.2004.04.016
- 4. Oncken C, Arias AJ, Feinn R, et al. Topiramate for Smoking Cessation: A Randomized, Placebo-Controlled Pilot Study. *Nicotine Tob Res.* 2014;16(3):288-296. doi:10.1093/ntr/ntt141
- 5. Dunn KE, Marcus TF, Kim C, Schroeder JR, Vandrey R, Umbricht A. Zonisamide Reduces Withdrawal Symptoms But Does Not Enhance Varenicline-Induced Smoking Cessation. *Nicotine Tob Res Off J Soc Res Nicotine Tob*. 2016;18(5):1171-1179. doi:10.1093/ntr/ntv236
- 6. Gadde KM, Yonish GM, Foust MS, Wagner HR. Combination therapy of zonisamide and bupropion for weight reduction in obese women: a preliminary, randomized, open-label study. *J Clin Psychiatry*. 2007;68(8):1226-1229. doi:10.4088/jcp.v68n0809
- 2010 Surgeon General's Report | Smoking & Tobacco Use | CDC.
   https://www.cdc.gov/tobacco/data\_statistics/sgr/2010/index.htm. Accessed March 2, 2020.
- 8. Jarvik M, Killen JD, Varady A, Fortmann SP. The favorite cigarette of the day. *J Behav Med*. 1993;16(4):413-422. doi:10.1007/BF00844781
- 9. Stahl SM, Pradko JF, Haight BR, Modell JG, Rockett CB, Learned-Coughlin S. A Review of the Neuropharmacology of Bupropion, a Dual Norepinephrine and Dopamine Reuptake Inhibitor. *Prim Care Companion J Clin Psychiatry*. 2004;6(4):159-166. doi:10.4088/pcc.v06n0403
- 10. Halo. https://www.halocigs.com/. Accessed February 26, 2020.
- 11. Gadde KM, Franciscy DM, Ii HRW, Krishnan KRR. Zonisamide for Weight Loss in Obese Adults: A Randomized Controlled Trial. *JAMA*. 2003;289(14):1820-1825. doi:10.1001/jama.289.14.1820
- 12. Wilkes S. The use of bupropion SR in cigarette smoking cessation. *Int J Chron Obstruct Pulmon Dis*. 2008;3(1):45-53.
- 13. Lee YY, Khoo S, Morris T, et al. A mixed-method study of the efficacy of physical activity consultation as an adjunct to standard smoking cessation treatment among male smokers in Malaysia. *SpringerPlus*. 2016;5(1):2012. doi:10.1186/s40064-016-3675-2
- 14. Zaccara G, Specchio LM. Long-term safety and effectiveness of zonisamide in the treatment of epilepsy: a review of the literature. *Neuropsychiatr Dis Treat*. 2009;5:249-259.

15. Fava M, Rush AJ, Thase ME, et al. 15 Years of Clinical Experience With Bupropion HCl: From Bupropion to Bupropion SR to Bupropion XL. *Prim Care Companion J Clin Psychiatry*. 2005;7(3):106-113.

Version 3.0 / 16 Feb 2021

16. Delnevo CD, Giovenco DP, Steinberg MB, et al. Patterns of Electronic Cigarette Use Among Adults in the United States. *Nicotine Tob Res Off J Soc Res Nicotine Tob*. 2016;18(5):715-719. doi:10.1093/ntr/ntv237
Appendix 1 - Patient Health Questionnaire (PHQ-9)

# PATIENT HEALTH QUESTIONNAIRE (PHQ-9)

Over the last 2 weeks, how often have you been bothered by any of the following problems?

| | Not at all | Several days | More than half<br>the days | Nearly every<br>day |
|---|---|---|---|---|
| 1. Little interest or pleasure in doing things | 0 | 0 | 0 | 0 |
| 2. Feeling down, depressed, or hopeless | 0 | 0 | 0 | 0 |
| 3. Trouble falling or staying asleep, or sleeping too much | 0 | 0 | 0 | 0 |
| 4. Feeling tired or having little energy | 0 | 0 | 0 | 0 |
| 5. Poor appetite or overeating | 0 | 0 | 0 | 0 |
| 6. Feeling bad about yourself- or that you are a failure or have let yourself or your family down | 0 | 0 | 0 | • |
| 7. Trouble concentrating on things, such as reading the newspaper or watching television | 0 | 0 | 0 | • |
| 8. Moving or speaking so slowly that other people could have noticed. Or the opposite- being so fidgety or restless that you have been moving around a lot more than usual | • | • | • | • |
| 9. Thoughts that you would be better off dead, or of hurting yourself in some way | 0 | 0 | 0 | • |

10. If you checked off any problems, how difficult have these problems made it for you to do your work, take care of things at home, or get along with other people?

- O Not difficult at all
- O Somewhat difficult
- O Very difficult
- O Extremely difficult

Appendix 2 – Fagerström Test for Nicotine Dependence (FTND)

# FAGERSTRÖM TEST FOR NICOTINE DEPENDENCE

INSTRUCTIONS: Please mark the answer that most accurately answers each question.

| I. F | low soon after you wake up | ob do | you smoke your first cigare | ette? | | | |
|---|---|---|---|---|---|---|---|
| 0 | Within 5 Minutes | 0 | 6-30 Minutes | 0 | 31-60 Minutes | 0 | After 60 Minutes |
| 2. [ | id you find it difficult to ref | rain | from smoking in places wh | ere i | t is forbidden, e.g., in churc | h, at | the library, in the cinema, etc.? |
| _ | Yes<br>No | | | | | | |
| 3. V | Vhich cigarette would you h | nate | most to give up? | | | | |
| 0 | The first one in the morn<br>Any other | ing | | | | | |
| 4. H | low many cigarettes per day | y do | you smoke? | | | | |
| 0 | 31 or more | 0 | 21-30 | 0 | 11-20 | 0 | 10 or less |
| 5. C | o you smoke more frequer | ntly o | during the first hours of wa | king | than during the rest of the | day? | ! |
| _ | Yes<br>No | | | | | | |
| 6. D | o you smoke if you are so | ill th | at you were in bed most of | the | day? | | |
| 0 | Yes<br>No | | | | | | |

Appendix 3 - Research Participant Payment Verification Form

### RESEARCH PARTICIPANT PAYMENT VERIFICATION FORM

#### **Receipt for Payment:**

In order for Rose Research Center to meet its obligations to the Internal Revenue Service we are required to obtain the following information. Payment received as compensation for participation in research is considered taxable income. You are responsible for paying any state, federal or Social Security taxes on the money you receive. If your total payment exceeds \$600 in any one calendar year, we are required to report this information to the Internal Revenue Service (IRS).

The Payment Verification Form will be used in order to process your payments only. Once your information has been entered into the Greenphire payment system, this form will be destroyed. Until that time, the form will be kept in a secure and locked area at all times. Your information will not be connected to your responses to the interviews, surveys, questionnaires or with your participation in this study.

| Full Name: | |
|-------------------------|------|
| Social Security Number: | |
| Permanent Home Address: | |
| · | <br> |
| | <br> |

### Appendix 4 – Smoking History

# **SMOKING HISTORY**

| What brand of c | igaret | ttes do you smoke? | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Color of cigarett | e pac | k? | | | | | | | | |
| Size: | 0 | Kings | O R | egu | lars O | 72's | 0 | 100's | 0 | 120's |
| Flavor: | 0 | Menthol | | o | Non-mentho | ol | | | | |
| Pack type: | О | Hard pack | | 0 | Soft pack | | | | | |
| Filtered? | О | Filtered | | 0 | Unfiltered | | | | | |
| I. How many ci | garet | tes do you smoke a day | ? | | | _cigs per day | | | | |
| 2. How old wer | e you | when you first smoked | a ciga | rett | e? | | years | old | | |
| 3. How old wer | How old were you when you became a regular smoker? years old | | | | | | | | | |
| 4. How many ye | ars h | ave you been a regular : | smoke | r? _ | | years | ; | | | |
| Have you beer<br>O Yes | n a re | gular smoker for the pas<br>O N | | ? | | | | | | |
| 5. How many ti | mes h | ave you tried to serious | ly quit | t sm | oking (for at I | east I day)?_ | | attempt | ts | |
| | | ed smoking, what was t | | | | e that you w | ere ab | le to stay off ci | garet | tes? (If less than 1 day, |
| O Hours | me si | eeping) O Days | | | O Weeks | | 1 C | Months | | O Years |
| 7. Have you part<br>O Yes | icipat | ed in a smoking study in<br>O N | | ast? | | | | | | |
| If YES, when | ? | | | ٧ | Where? | | | | _ | |
| 8. Are you inter<br>O Yes | ested | I in switching from a cor<br>O N | | ble | cigarette to ai | n electronic o | igaret | te? | | |
| 9. Have you smo<br>O Yes | oked | cigar in the past 14 days<br>O No | | | | | | | | |
| 10. Have you sm<br>O Yes | oked | a pipe, hookah or an e-<br>O No | | tte i | n the past 14 | days? | | | | |
| II. Have you us<br>O Yes | ed sn | uff or chewing tobacco<br>O No | | pas | t 14 days? | | | | | |

# Appendix 5 – Registration Form

### REGISTRATION FORM

(Please Print)

| | | | COI | NTACT IN | IFORM | IATIO | DN | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Last Name: | | | | First: | | | ١ | fiddle Initial: | ☐ Mr.<br>☐ Mrs. | ☐ Miss<br>☐ Ms. |
| Street Address: | | | | | | | | | | , |
| P.O. Box: | City: State: | | | | | | | ZIP Code: | | |
| E-mail Address: | | | | | | | Do you have w | eb access othe | | - |
| | | | | | | | | | □ Yes | □ No |
| Primary Phone Nur | nary Phone Number: Cell Other Phone Number: Office Home ( ) | | | | | | | | | Cell<br>Office<br>Home |
| Do you give Rose f | Research Cen | ter permission to | | | ove numb | ers? | | | ☐ Yes | □ No |
| Emergency contact: | | | | | | | with: | | | |
| Name of local frien | | | | Relationship | | - | Phone no.: | | | |
| | | | | - | | | ( ) | | | |
| (Initial here) | , , | | | | | | | | | |
| DEMOGRAPHIC INFORMATION | | | | | | | | | | |
| Birth Date: / | | Sex: 🗆 M | | Marital Sta | | | Single / Marrie | ed / Divorced | d / Separated | / Widowed |
| Race: Ethnicity: American Indian or Alaska Native Hispanic or Latino Not Hispanic or Latino | | | | | | | | | | |
| Are you a U.S. Vet | eran? | | | | | | | | ☐ Yes | □No |
| Are you currently | employed at o | r have affiliation v | vith the Ro | se Research C | enter? | | | | □ Yes | □No |
| Are you currently | participating in | another clinical ( | trial? | | | | | | □ Yes | □No |
| Have you participal | ted in a clinica | l trial in the past : | 3 months t | hat included an | investigati | tional dru | ug? | | □ Yes | □No |
| I attest that all of the information above is to the best of my knowledge and believe true, correct and complete. | | | | | | | | | | |
| | Partici | pant's Signature | | | | | | Date | | |
| | | I | DENTI | FICATIO | | IFICA | TION | | | |
| | Form | of ID Verified: | ☐ Drive | | use only) | o ID ( | □ Military ID | ☐ Passpo | rt | |
| | Research F | ersonnel's Signati | ıre | | | | | Date | | |

Appendix 6 – Medical History Form

# MEDICAL HISTORY FORM

| Major | Medica | I Conditions |
|---|---|---|
| | L | -d |
| ☐ Yes | □ No | ad or are currently having/ being treated for any of the following conditions? High blood pressure (Hypertension) |
| Yes | □ No | Heart attack, Heart Failure, OR heart disease diagnosis by cardiac angiogram |
| ☐ Yes | □ No | Problems with heart valves such as mitral regurgitation, stenosis, artificial valve or other |
| Yes | □ No | |
| Yes | □ No | Heart rhythm problem such as atrial fibrillation, tachycardia, or pacemaker |
| Yes | □ No | Prior surgery on the gastrointestinal tract (e.g. colectomy, gastric by-pass, Reux-En-Y) Skin problems |
| ☐ Yes | □ No | Cirrhosis of the liver |
| ☐ Yes | □ No | Liver problems other than cirrhosis (e.g. Hepatitis, fatty liver) |
| Yes | □ No | Kidney failure |
| Yes | □ No | Chronic Kidney Disease |
| Yes | □ No | Chronic Diarrhea and/or constipation such as Irritable Bowel Syndrome, Crohn's Disease, Inflammatory Bowel |
| Yes | □ No | Stomach/ Duodenal Ulcer (Gastrointestinal Ulcer) |
| Yes | □ No | Chronic Bronchitis (cough every morning) |
| Yes | □ No | Chronic Obstructive Pulmonary Disease (COPD) or Emphysema |
| Yes | □ No | Other lung disorder such as Tuberculosis, Pulmonary Fibrosis, Sarcoid |
| Yes | □ No | Asthma |
| Yes | □ No | Stroke or TIA (mini stroke) |
| Yes | □ No | Seizure/ epilepsy |
| Yes | □ No | Migraine headaches |
| Yes | □ No | Unexplained fainting spells |
| ☐ Yes | □ No | Insomnia |
| ☐ Yes | □ No | Other neurologic conditions |
| ☐ Yes | □ No | Problems giving blood samples |
| ☐ Yes | □ No | Anemia requiring iron |
| ☐ Yes | □ No | Blood disorder |
| ☐ Yes | □ No | Rheumatic Disease such as Rheumatoid Arthritis, Fibromyalgia, other |
| ☐ Yes | □ No | Sinusitis/ Seasonal allergies |
| ☐ Yes | □ No | Other severe allergies |
| ☐ Yes | □ No | Diabetes or Pre-diabetes |
| ☐ Yes | □ No | Thyroid disease or condition |
| ☐ Yes | □ No | Cancer |
| ☐ Yes | □ No | Depression/ Anxiety/ Bipolar disorder |
| ☐ Yes | □ No | Post-traumatic stress disorder |
| ☐ Yes | □ No | Other Psychiatric problems (e.g., Borderline, Schizoaffective, Schizophrenia, Hypomania, ADHD) |
| ☐ Yes | □ No | History of Sexually Transmitted Disease (STD) |
| ☐ Yes | □ No | Chronic infectious syndrome such as HIV, CMV, Epstein Barr |
| ☐ Yes | □ No | History of drug or alcohol abuse |
| ☐ Yes | □ No | Intolerance to medications |
| ☐ Yes | □ No | Other major medical condition |

| Office use only: |
|------------------|

| Past | t Medical History | |
|---|---|---|
| Pleas | e list any illnesses that have caused you to miss work or have interrupted your life this past year: | |
| I. | | Mo/Yr: |
| 2. | | Mo/Yr: |
| 3. | | Mo/Yr: |
| 4. | | Mo/Yr: |
| 5. | | Mo/Yr: |
| Pleas | e list any hospitalizations. If possible, include the year: | |
| I. | | Mo/Yr: |
| 2. | | Mo/Yr: |
| 3. | | Mo/Yr: |
| 4. | | Mo/Yr: |
| 5. | | Mo/Yr: |
| Pleas | e list any serious injuries or accidents. If possible, include the year: | |
| I. | | Mo/Yr: |
| 2. | | Mo∕Yr: |
| 3. | | Mo/Yr: |
| 4. | | Mo/Yr: |
| 5. | | Mo/Yr: |
| Pleas | e list any surgeries or major procedures, along with the reason. If possible, include the year: | |
| I. | | Mo/Yr: |
| 2. | | Mo/Yr: |
| 3. | | Mo/Yr: |
| 4. | | Mo/Yr: |
| 5. | | Mo/Yr: |
| | Office use only: | |

Page 2 of 5

| Family History Please mark an "x" for any first-degree family member(s) (children, parents, or siblings) that currently has or had any of the following | | | | | | | |
|---|---|---|---|---|---|---|---|
| Please mark an "x" for any first-degree family member<br>illnesses (select all that apply): | er(s) (childre | n, parents | , or siblings) th | nat currently | has or had an | y of the foll | owing |
| llness | Mother | Father | Sister | Brother | Daughter | Son | None |
| Anemia or Blood disease | | | oister . | | | | |
| Cancer | | _ | _ | _ | _ | _ | _ |
| Diabetes | _ | _ | _ | _ | _ | _ | _ |
| Glaucoma | | | | | | | |
| Heart disease | | | | | | | |
| High blood pressure | | | | | | | |
| Mental Illness/ Depression/ Generalized Anxiety | | | | | | | |
| Stroke | | | | | | | |
| Substance abuse (alcohol, tobacco or other) | | | | | | | |
| Other serious illness: | | | | | | | |
| Social History | | | | | | | |
| Please complete the following questions: | | | | | | | |
| Do you drink alcohol, beer, or wine? | ☐ Yes | □ No | If YES, how r | nany drinks į | er week? | | |
| | | | How many d<br>of the week? | | have on your | heaviest dr | inking day |
| Do you drink coffee, tea, caffeinated soda daily? | ☐ Yes | □ No | If YES, how r | nany cups pe | er day? | | |
| Have you used a non-prescription drug such as marijuana, cocaine, heroin in the last month? Have you used prescription drugs not prescribed to you? | ☐ Yes | □ No | If YES, when | and what dr | ug/ substance : | and last dat | e of use: |
| Have you used an Experimental (investigational) drug<br>or biologic in the past 30 days? | Yes 🗅 Yes | □ No | | | | | |
| Blood Donation | | | | | | | |
| Please complete the following question: | | | | | | | |
| Have you donated any blood or blood products within the last 2 months? | ☐ Yes | □ No | If YES, what letc.)? | blood produ | ct (whole bloo | od, plasma, p | olatelets, |
| General Health | | | | | | | |
| Please complete the following questions: | | | | | | | |
| Do you use supplemental oxygen? | | □ No | | | | | |
| Can you walk up 2 flights of stairs? | , without sto | pping [ | Yes, but I ne | ed to stop a | long the way | □ No | |

| General Health (conti | inued) | | | | | |
|---|---|---|---|---|---|---|
| How well do you walk? | | ☐ Independent | y 🔲 I use a cane | or walker | ☐ I use a w | heelchair |
| Do you use CPAP machine? | | ☐ Yes | □ No | | | |
| General Health (Won | nen Only) | | | | | |
| Do you agree to use a medical of the study? | lly acceptable fo | orm of birth con | trol for the duration | | □ Y | es 🚨 No |
| If yes, please select form of co | ntraception you | and/or your pa | rtner plan to use or | are currently u | ısing. | |
| ☐ Tubal ligation / Hysterecton | ny / Bilateral oo | phorectomy | ☐ Vasector | my | | |
| ☐ Birth control pills / patches | / implants / inje | ections | ☐ Not het | erosexually ac | tive | |
| ☐ Condom / Diaphragm used | with spermicid | e | ☐ None | | | |
| ☐ Intrauterine device (IUD) / | Essure | | ☐ Post-m | enopausal | | |
| Medications | | | | | | |
| Please list any allergies and the | reaction cause | d by the allergy | (e.g. "rash" or "tong | ue swelling" or | "itchiness"): | |
| Trease including and great arise and | | o by the anergy | (1.2. 1231 51 551) | | 10011111020 / | |
| Medications List Please list all medications you prescriptions): | Please list all medications you have used within the last month (include over-the counter drugs, vitamins/ supplements, and especially | | | | | |
| Name of medication | Dosing (mg/t<br>Route (oral, | | Frequency<br>(times per day) | Start date | Stop date | Prescribed for what problem? |

| Smoking Cessation Products | | | | | |
|---|---|---|---|---|---|
| For each of the following, mark if you have used the product, experienced any side effects, allergy or intolerance with usage or had to | | | | | |
| stop using the product due to side effects: | | | | | |
| | | | | Stopped | |
| | Not Used | Used | Side Effects | Side Effec | _ |
| Nicotine Patch | | | | □ Yes | ☐ No |
| Nicotine Gum | | | | ☐ Yes | □ No |
| Nicotine Lozenge | | | | ☐ Yes | □ No |
| Nicotine Inhaler | | | | ☐ Yes | □ No |
| Nicotine Nasal Spray | | | | ☐ Yes | □ No |
| Zyban (wellbutrin) | | | | ☐ Yes | □ No |
| Chantix (varenicline) | | | | ☐ Yes | □ No |
| Have you used any of these products within the past 14 days? | | | | | |

| MD/ PA Signature | Date |
|------------------|------|

Page 5 of 5

Appendix 7- Review of Systems Form

### **REVIEW OF SYSTEMS**

| Are you currently (in the last 30 days) ha | ving/ being treated for any of the followi | ng conditions: |
|---|---|---|
| General: ( none of these apply) Unexplained weight loss or gain Fatigue/ Lack of energy | ☐ Fever or chills☐ Weakness | ☐ Trouble Sleeping |
| Skin: ( none of these apply) Rashes Lumps | ☐ Itching ☐ Dryness | ☐ Color changes☐ Hair and nail changes |
| Head: ( none of these opply) Headache | ☐ Head Injury | |
| Ears: ( none of these opply) Decreased hearing | ☐ Earache | ☐ Ringing in ears |
| Eyes: ( none of these apply) Vision problems Specks | ☐ Blurry or double vision☐ Flashing lights | ☐ Redness<br>☐ Pain |
| Nose: ( none of these apply) ☐ Stuffiness ☐ Discharge | ☐ Itching☐ Sinus pain | ☐ Nose Bleeds |
| Throat: ( none of these opply) Teeth/gum problems Dentures Hoarseness | □ Sore tongue □ Dry mouth □ Sore throat | ☐ Thrush☐ Non-healing sores☐ Difficulty swallowing |
| Neck: ( none of these opply) □ Lumps □ Stiffness | ☐ Pain | ☐ Swollen glands |
| Respiratory: ( none of these opply) Cough (dry or wet, productive) Shortness of breath | ☐ Coughing up blood☐ Painful breathing | ☐ Wheezing |
| Cardiovascular: ( none of these opply) Chest pain or discomfort Tightness Heart pounding/ Fluttering/ Palpitations | ☐ Difficulty breathing lying down ☐ Swelling ☐ Shortness of breath with activity | ☐ Suddenly awaking from sleep with shortness of breath |
| Gastrointestinal: ( none of these opply) □ Swallowing difficulties □ Heartburn □ Constipation □ Vomiting | ☐ Change in bowel habits ☐ Rectal bleeding ☐ Diarrhea ☐ Stomach pain | ☐ Yellow eyes or skin☐ Change in appetite☐ Nausea |
| Urinary: ( none of these opply) ☐ Frequency ☐ Urgency | ☐ Blood in urine☐ Pain with urination | ☐ Change in urinary strength☐ Incontinence |

### REVIEW OF SYSTEMS

| () Leg cramping Leg pains |
|------------------------------------------------------|
| Back pain Swelling of joints Trauma |
| Depty) Weakness Numbness Shaking episodes |
| opply) □ Bleed easily |
| ply) Frequent urination Change in appetite Thirst |
| pply) Memory loss Feeling down |
| арр(у)<br>eeding |
| Office Use Only |
| Date Date |
| Weakness Tremor Shaking episodes |

Appendix 8 – Employment History

### **EMPLOYMENT HISTORY**

| ١. | Wha | t is the highest degree you have completed? |
|---|---|---|
| | 0 0 0 0 0 | High school diploma or G.E.D. Technical degree Two year associates degree (e.g. A.A.) Four year undergraduate degree (e.g. B.A., B.S.) Professional degree (e.g. P.A., R.N.) Master's degree (e.g. M.A., M.S., M.B.A.) Doctorate (e.g. Ph. D., M.D., J.D.) Other |
| 2. | How | many years of formal education have you completed: (Include grade school and higher) |
| 3. | Wha | t is your current employment status? |
| | 0 | Not employed (please answer question 4) Part-Time work Full-time work |
| 4. | If not | t employed is selected, please specify your answer: |
| | 0 0 0 | Education (Full-time student) Retired Medical leave Homemaker Laid off Other |
| 5. | Wha | t is your current job title; if no longer employed, in what position were you last employed? |
| 6. | How | physically demanding is your current employment? |
| 000 | Ver<br>A li | t employed t demanding at all y little demanding ttle demanding newhat demanding derately demanding |
| | | y demanding |

| 7. | How mentally or emotionally stressful is your current employment? |
|---|---|
| 0 | Not employed |
| $\circ$ | Not stressful at all |
| $\circ$ | Very little stress |
| $\circ$ | A little stressful |
| $\circ$ | Somewhat stressful |
| $\circ$ | Moderately stressful |
| $\circ$ | Very stressful |
| 0 | Extremely stressful |
| 8. | What is your gross (before taxes) annual household income? |
| 0 | < \$16,000 |
| 0 | \$16,001- \$32,000 |
| $\circ$ | \$32,001- \$48,000 |
| О | \$48,001-\$64,000 |
| 0 | \$64,001-\$80,000 |
| $^{\circ}$ | \$80,001- \$96,000 |
| 0 | >\$96,000 |
| 9. | What are your estimated total assets? (Include house, automobiles, stocks, savings, furniture, etc.). |
| 0 | <\$50,000 |
| О | \$50,001-\$100,000 |
| О | \$100,001-\$200,000 |
| 0 | \$200,001- \$300,000 |
| $\circ$ | \$300,001- \$400,000 |
| $^{\circ}$ | \$400,001- \$500,000 |
| 0 | \$500,001- \$750,000 |
| 0 | >\$750,001 |
| 10. | How many people live in your household? |

Appendix 9 – modified Cigarette Evaluation Questionnaire - Ext (mCEQ-E)

# CIGARETTE EVALUATION QUESTIONNAIRE- Ext modified

Have you smoked any cigarettes since your last visit?

- O No: Skip questionnaire
- O Yes: Please answer the following questions based on the **FIRST** cigarette you smoked on the last day you smoked.

| | Not<br>at all | Very<br>little | A<br>little | Moderately | A lot | Quite a<br>lot | Extremely |
|---|---|---|---|---|---|---|---|
| 1. Was it satisfying? | 0 | 0 | О | 0 | 0 | 0 | 0 |
| 2. Did it taste good? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 3. Did it make you dizzy? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 4. Did it calm you down? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 5. Did it help you concentrate? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 6. Did it make you feel more awake? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 7. Did it reduce your hunger for food? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 8. Did it make you nauseated? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 9. Did it make you feel less irritable? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 10. Did you enjoy the sensations of the smoke in your throat and chest? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| II. Did it immediately reduce your craving for cigarettes? | 0 | 0 | o | 0 | 0 | 0 | o |
| 12. Did you enjoy smoking? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |

#### Please answer the following questions based on the cigarette smoked immediately after a meal.

O Did not smoke immediately after a meal: Skip section

| | Not at<br>all | Very<br>little | A<br>little | Moderately | A lot | Quite a<br>lot | Extremely |
|---|---|---|---|---|---|---|---|
| 1. Was it satisfying? | 0 | O | 0 | 0 | О | 0 | 0 |
| 2. Did it taste good? | 0 | 0 | 0 | 0 | O | 0 | 0 |
| 3. Did it make you dizzy? | 0 | 0 | 0 | 0 | O | 0 | 0 |
| 4. Did it calm you down? | 0 | 0 | 0 | 0 | O | 0 | 0 |
| 5. Did it help you concentrate? | 0 | 0 | 0 | 0 | O | 0 | 0 |
| 6. Did it make you feel more awake? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 7. Did it reduce your hunger for food? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 8. Did it make you feel nauseated? | 0 | 0 | 0 | 0 | O | 0 | 0 |
| 9. Did it make you feel less irritable? | 0 | 0 | 0 | 0 | o | 0 | O |

| 10. Did you enjoy the sensations of the smoke in<br>your throat and chest? | o | О | o | o | 0 | 0 | 0 |
|---|---|---|---|---|---|---|---|
| II. Did it immediately reduce your craving for cigarettes? | o | o | 0 | o | 0 | 0 | 0 |
| 12. Did you enjoy smoking? | 0 | O | 0 | 0 | O | 0 | 0 |

Please answer the following questions regarding all other cigarettes smoked on the last day you smoked.

| ricase answer are following questions regarding an e | | | | | , , | | |
|---|---|---|---|---|---|---|---|
| | Not<br>at all | Very<br>little | A<br>little | Moderately | A lot | Quite a<br>lot | Extremely |
| 1. Was it satisfying? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 2. Did it taste good? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 3. Did it make you dizzy? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 4. Did it calm you down? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 5. Did it help you concentrate? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 6. Did it make you feel more awake? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 7. Did it reduce your hunger for food? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 8. Did it make you nauseated? | 0 | O | 0 | 0 | 0 | 0 | 0 |
| 9. Did it make you feel less irritable? | 0 | O | 0 | 0 | 0 | 0 | 0 |
| 10. Did you enjoy the sensations of the smoke in your throat and chest? | o | o | 0 | 0 | 0 | 0 | 0 |
| 11. Did it immediately reduce your craving for cigarettes? | o | o | o | 0 | 0 | 0 | 0 |
| 12. Did you enjoy smoking? | 0 | О | 0 | 0 | 0 | 0 | 0 |

Appendix 10 – modified Electronic Cigarette Evaluation Questionnaire - Ext (mECEQ-E)

### ELECTRONIC CIGARETTE EVALUATION QUESTIONNAIRE- Ext modified

Have you used any ELECTRONIC cigarettes since your last visit?

- O No: Skip questionnaire
- O Yes: Please answer the following questions based on the **FIRST** use of the day on the last day you used the <u>ELECTRONIC</u> cigarette.

| <u>=====================================</u> | | | | | | | |
|---|---|---|---|---|---|---|---|
| | Not<br>at all | Very<br>little | A<br>little | Moderately | A lot | Quite a<br>lot | Extremely |
| 1. Was it satisfying? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 2. Did it taste good? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 3. Did it make you dizzy? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 4. Did it calm you down? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 5. Did it help you concentrate? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 6. Did it make you feel more awake? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 7. Did it reduce your hunger for food? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 8. Did it make you nauseated? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 9. Did it make you feel less irritable? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 10. Did you enjoy the sensations of the smoke in<br>your throat and chest? | o | 0 | 0 | 0 | 0 | o | 0 |
| II. Did it immediately reduce your craving for cigarettes? | 0 | 0 | 0 | 0 | 0 | o | 0 |
| 12. Did you enjoy smoking? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |

#### Please answer the following questions based on the use of the ELECTRONIC cigarette immediately after a meal.

O Did not use the ELECTRONIC cigarette immediately after a meal: Skip section

| | Not at<br>all | Very<br>little | A<br>little | Moderately | A lot | Quite a<br>lot | Extremely |
|---|---|---|---|---|---|---|---|
| 1. Was it satisfying? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 2. Did it taste good? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 3. Did it make you dizzy? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 4. Did it calm you down? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 5. Did it help you concentrate? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 6. Did it make you feel more awake? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 7. Did it reduce your hunger for food? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 8. Did it make you feel nauseated? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 9. Did it make you feel less irritable? | 0 | 0 | 0 | 0 | 0 | 0 | O |

| 10. Did you enjoy the sensations of the smoke in<br>your throat and chest? | o | o | o | 0 | O | 0 | 0 |
|---|---|---|---|---|---|---|---|
| II. Did it immediately reduce your craving for cigarettes? | o | o | o | o | 0 | 0 | 0 |
| 12. Did you enjoy smoking? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |

Please answer the following questions regarding <u>all other times you used the ELECTRONIC cigarette</u> on the last day you used the ELECTRONIC cigarette.

| | Not<br>at all | Very<br>little | A<br>little | Moderately | A lot | Quite a<br>lot | Extremely |
|---|---|---|---|---|---|---|---|
| 1. Was it satisfying? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 2. Did it taste good? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 3. Did it make you dizzy? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 4. Did it calm you down? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 5. Did it help you concentrate? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 6. Did it make you feel more awake? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 7. Did it reduce your hunger for food? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 8. Did it make you nauseated? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 9. Did it make you feel less irritable? | 0 | О | 0 | 0 | O | 0 | 0 |
| 10. Did you enjoy the sensations of the smoke in your throat and chest? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| II. Did it immediately reduce your craving for cigarettes? | 0 | o | o | 0 | 0 | o | 0 |
| 12. Did you enjoy smoking? | 0 | 0 | 0 | 0 | O | 0 | 0 |

Appendix 11 – Halo G6 Flavor Assessment Questionnaire

### **HALO G6 Flavor Assessment Questionnaire**

Now that you have tried the two flavors of HALO G6, are you willing to switch to either of these flavors?

(CHECK ONE RESPONSE ONLY)

YES\_\_\_\_\_\_\_ No\_\_\_\_\_

If YES, which flavor would you like to use:

Tribeca (tobacco)\_\_\_\_\_\_ Mint\_\_\_\_\_

Participant's Signature and Date

Appendix 12 - Participant Instructions for Varenicline



### INSTRUCTIONS FOR PROPER USE OF BUPROPION (ZYBAN)

#### How does it work?

This medicine helps a person to stop smoking by reducing the desire (urge) to smoke.

#### How do I take this medicine?

- 1. Take bupropion exactly as directed. The blister packs are designed to help you take the medicine properly.
  - a. For the first 3 days, take one tablet (150 mg) in the morning.
  - b. For the rest of the time, take two tablets (150 mg  $\times$  2) in the morning.
  - c. Only change your medicine at the direction of the study personnel or if you have a serious concern.
- 2. Do not crush, chew or split the tablet
- Take bupropion with a full glass (8 ounces) of water. You may take bupropion with or without food (do NOT drink alcohol with bupropion).
- We will schedule you to start taking bupropion about 7 days before your actual switch date (the day you stop smoking and only use electronic cigarettes).
- If you forget to take a dose of bupropion, take is as soon as you remember. If it is almost time for your next dose (less than 6 hours), just wait and take your next dose at the regular time. Do NOT take an extra dose to make up for the dose you forgot.
- Keep this medication in a safe place, AWAY FROM CHILDREN. It should be stored at room temperature (not in your car) and away from direct sun, excessive heat, cold, or moisture. You MUST return any unused medication.

#### Precautions

Some people have reported changes in behavior, agitation, depression, thoughts of suicide, or hostility. If you experience any of these issues, please call Rose Research Center and speak with one of our helpful staff (919-328-2345). You may also call the 24-hour emergency advice line and speak with our study physician (855-999-1940) if you feel this is an emergency.

As with most any medication, there is a risk of having an allergic reaction to bupropion. This can be serious, especially if you experience swelling of the face, mouth, tongue, or throat which causes difficulty breathing. If you have any of these symptoms, stop taking bupropion and get medical attention right away. Inform the staff at Rose Research Center AFTER you obtain medical care for these symptoms.

You should tell the staff at Rose Research Center if you have any allergies to medicines, including bupropion.

You should also inform the staff at Rose Research Center if you believe you may be pregnant (for women only).

Use caution driving and operating machinery when you first start taking bupropion until you know how it is going to affect you. Some people feel dizzy or have trouble concentrating when they first start bupropion.

#### Potential Side Effects

In some people, bupropion can cause:

| Dry mouth | Insomnia (trouble sleeping) |
|------------------------------|-----------------------------|
| Unusual dreams | Mood changes |
| Headaches | Constipation (hard to poop) |
| Change in appetite or weight | Excitement or anxiety |

If you experience any of these side effects, or any other side effects, please notify the staff at Rose Research Center.

Appendix 13 – Participant Instructions for Zonisamide



### INSTRUCTIONS FOR PROPER USE OF ZONISAMIDE (ZONEGRAN)

#### How does it work?

This medicine is normally used to prevent seizures, but it may help with switching to sole use of an electronic cigarette.

#### How do I take this medicine?

- 1. Take zonisamide exactly as directed. The blister packs are designed to help you take the medicine properly.
  - Take 2 capsules (50 mg each, total of 100 mg) in the morning.
  - b. Only change your medicine at the direction of the study personnel or if you have a serious concern.
- Do not take this medicine if you have a severe allergy to sulfa drugs (like Bactrim, Septra, Diabeta).
- 3. Do not crush, chew, open or split the capsule.
- Take zonisamide with a full glass (8 ounces) of water. Zonisamide can be taken with or without food (do NOT drink alcohol with zonisamide).
- We will schedule you to start taking zonisamide about 7 days before your actual switch date (the day you stop smoking and only use the electronic cigarette).
- If you forget to take a dose of zonisamide, take is as soon as you remember. If it is almost time for your next dose (less than 6 hours), just wait and take your next dose at the regular time. Do NOT take an extra dose to make up for the dose you forgot.
- Keep this medication in a safe place, AWAY FROM CHILDREN. It should be stored at room temperature (not in your car) and away from direct sun, excessive heat, cold, or moisture. You MUST return any unused medication.

#### Precautions

Some people have reported changes in behavior, agitation, depression, thoughts of suicide, or hostility. If you experience any of these issues, please call Rose Research Center and speak with one of our helpful staff (919-328-2345). You may also call the 24-hour emergency advice line and speak with our study physician (855-999-1940) if you feel this is an emergency.

As with most any medication, there is a risk of having an allergic reaction to zonisamide. This can be serious, especially if you experience swelling of the face, mouth, tongue, or throat which causes difficulty breathing. If you have any of these symptoms, stop taking zonisamide and get medical attention right away. Inform the staff at Rose Research Center AFTER you obtain medical care for these symptoms.

You should tell the staff at Rose Research Center if you have any allergies to medicines, including zonisamide or sulfadrues.

You should also inform the staff at Rose Research Center if you believe you may be pregnant (for women only).

Use caution driving and operating machinery when you first start taking zonisamide until you know how it is going to affect you. Some people feel sleepy, dizzy, or have trouble concentrating when they first start zonisamide.

#### Potential Side Effects

In some people, zonisamide can cause:

| Nausea (feel like throwing up) | Drowsiness |
|--------------------------------|-----------------------------|
| Dizziness | Heartburn |
| Headaches | Constipation (hard to poop) |
| Weight loss | Dry mouth |

If you experience any of these side effects, or any other side effects, please notify the staff at Rose Research Center.

Appendix 14 – Assessment of Behavioral OUTcomes (ABOUT)

#### ASSESSMENT of BEHAVIORAL OUTcomes (ABOUT)

#### Related to Tobacco and nicotine products

The next questions ask about your experience with tobacco and nicotine products. Please answer all questions. Please think about all the tobacco and nicotine products that you use as you answer all of the following questions.

1. Over the past 7 days, on average, how soon after you woke up did you use your first product?

| 0 to 5 minutes |
|-----------------------------|
| 6 to 15 minutes |
| 16 to 30 minutes |
| 31 to 60 minutes |
| More than 1 hour to 3 hours |
| More than 3 hours |

2. Over the past 7 days, on average, how long before going to sleep did you use your last product?

| 0 to 5 minutes |
|-----------------------------|
| 6 to 15 minutes |
| 16 to 30 minutes |
| 31 to 60 minutes |
| More than I hour to 3 hours |
| More than 3 hours |

# ASSESSMENT of BEHAVIORAL OUTcomes (ABOUT)

### Related to Tobacco and nicotine products

| 3. Currently | Not at all | A little | Moderately | Very Much | Extremely |
|---|---|---|---|---|---|
| a. How much do you feel you need<br>your product(s) to function<br>"normally"? | 0 | 0 | 0 | 0 | 0 |
| How difficult do you think it would be for you to completely quit your product(s)? | 0 | 0 | 0 | 0 | 0 |

| 4. Over the past 7 days, how often did you | Never | Rarely | Sometimes | Most of the time | All the time |
|---|---|---|---|---|---|
| a. Have a strong desire to use your product(s)? | o | 0 | 0 | 0 | 0 |
| b. Use more of your product(s) than you intend to? | 0 | 0 | 0 | 0 | 0 |
| c. Feel that you "HAD to have one"? | 0 | 0 | 0 | 0 | 0 |
| d. Use your product(s) in a situation where you weren't supposed to? | o | 0 | 0 | 0 | 0 |
| e. Find it hard to control the need or urge to use your product(s)? | 0 | 0 | 0 | 0 | 0 |
| f. Sneak off to use your product(s)? | 0 | 0 | 0 | 0 | 0 |
| g. Avoid an activity because you couldn't use your product(s)? | 0 | 0 | 0 | 0 | 0 |
| h. Stop what you were doing to use your product(s)? | 0 | o | 0 | 0 | 0 |

#### Appendix 15 - Session Payment Form

For your time and inconvenience related to your participation in this study, you will be paid up to a total of \$950 if you complete this study. If you do not complete the study, for any reason, you will be paid for the study visits you do complete according to the following schedule:

- · You will receive \$25 for completing Study Visit 1.
- You will receive \$75 for completing Study Visit 2 through Study Visit 7 (\$450 total)
- You will receive \$5 for responding to each text message during the study (once per day for approximately 91 - 95 days = approximately \$475). In order to receive compensation for each message, you will need to answer all of questions before you receive your next text message.

#### SESSION PAYMENT LOG

| | DATE | AMOUNT ELIGIBLE | AMOUNT ELIGIBLE | AMOUNT TO | RRC | PARTICIPANT | DATE |
|---|---|---|---|---|---|---|---|
| SESSION | ATTENDED | VISIT | SMS | BE PAID | INITIALS | INITIALS | PROCESSED |
| Visit 1-Screen | | \$25 | \$0 | | | | |
| Visit 2 | | \$75 | \$0 | | | | |
| SMS | | | x \$5 | | | | |
| Visit 3 | | \$75 | | | | | |
| SMS | | | x \$5 | | | | |
| Visit 4 | | \$75 | | | | | |
| SMS | | | x \$5 | | | | |
| Visit 5 | | \$75 | | | | | |
| SMS | | | x \$5 | | | | |
| Visit 6 | | \$75 | | | | | |
| SMS | | | x \$5 | | | | |
| Visit 7 | | \$75 | | | | | |
| SMS | | | x \$5 | | | | |
| TOTAL | | \$475 | | | | | |

I certify that the payment eligibility process has been fully explained to me and I agree with and accept all conditions of the payment eligibility process.

| Date |
|------|
| Date |

Appendix 16 – Reasons to Smoke

#### **REASONS TO SMOKE**

Version 3.0 / 16 Feb 2021

Have you smoked any cigarettes since your switch day?

- O No: Skip questionnaire
- O Yes: Please answer the following questions based on the FIRST cigarette you smoked on the last day you smoked.

INSTRUCTIONS: Listed below are thirteen common reasons why people like to smoke. Using the scale on the right, fill in the bubble for each statement which most closely describes how important that reason is to you.

| | Least<br>Important | Hardly<br>Important | Not Really<br>Important | A Little<br>Important | More<br>Important | Really<br>Important | Most<br>Important |
|---|---|---|---|---|---|---|---|
| I. It calms me down | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 2. It gives me something to do with my hands | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 3. I like the taste and smell | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 4. I like the sensations deep in my throat or chest | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 5. It wakes me up when I am drowsy | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 6. I like to watch the smoke | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 7. It makes relaxing seem even better | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 8. It satisfies my craving | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 9. It gives me a rush | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 10. It gives me more confidence around other people | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| II. It helps me control my weight | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 12. It's is like a friend | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 13. It helps me concentrate | 0 | 0 | 0 | 0 | 0 | 0 | 0 |

Appendix 17 – Shiffman Jarvik Withdrawal Scale

# SHIFFMAN-JARVIK WITHDRAWAL SCALE

INSTRUCTIONS: Please fill in the bubble for each question that most accurately reflects how you have felt TODAY.

| | Not at all | Very little | A little | Moderately | A lot | Quite a lot | Extremely |
|---|---|---|---|---|---|---|---|
| If you could have smoked freely,<br>would you have liked a cigarette?<br>(your own brand) | 0 | 0 | 0 | 0 | 0 | 0 | o |
| Has your heart beat faster than usual? | 0 | 0 | 0 | 0 | 0 | 0 | o |
| Have you felt more calm than usual? | 0 | 0 | 0 | 0 | 0 | 0 | o |
| Have you been able to concentrate? | 0 | o | 0 | 0 | 0 | 0 | o |
| Have you felt wide awake? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Have you felt content? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Have you thought of cigarettes?<br>(your own brand) | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Have you had fluttery feelings in your chest? | 0 | o | 0 | 0 | 0 | 0 | o |
| Have you felt hungrier than usual? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| If you were permitted to smoke,<br>how likely is it that you would<br>have refused a cigarette? (your<br>own brand) | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Have you felt tense? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Have you missed smoking a cigarette? (your own brand) | 0 | 0 | 0 | 0 | 0 | 0 | o |
| Do you have the urge to smoke a cigarette? (your own brand) | 0 | 0 | 0 | 0 | 0 | 0 | o |
| Have you felt irritable? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Have your hands been shaky? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Have you eaten more than usual? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Have you missed something to do with your hands? | 0 | o | 0 | 0 | 0 | 0 | o |
| Have you missed having something in your mouth? | 0 | o | 0 | o | 0 | 0 | o |

| | Not at all | Very little | A little | Moderately | A lot | Quite a lot | Extremely |
|---|---|---|---|---|---|---|---|
| Did you have trouble sleeping last night? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Have you had a headache? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Have you had an upset stomach? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Have you felt dizzy? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Have you had a bad taste in your mouth? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Have you had a cough? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Have you had mouth sores? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Have you felt nauseated? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Have you had a sore throat? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Have you craved sweets? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Have you had heartburn? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Have you craved salty foods? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Have you felt a tightness in your chest? | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Have you craved a cigarette? (your own brand) | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Have you missed inhaling cigarette smoke? | o | o | 0 | o | 0 | 0 | 0 |